CLINICAL TRIAL: NCT01149369
Title: Aprepitant for the Relief of Nausea in Patients With Chronic Nausea and Vomiting of Presumed Gastric Origin: A Multicenter, Randomized, Double-Masked, Placebo-Controlled Trial
Brief Title: Aprepitant for the Relief of Nausea in Patients With Chronic Nausea and Vomiting of Presumed Gastric Origin Trial
Acronym: APRON
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IND - DK-GpCRC-4APRON; U01DK073983 (NIH); U01DK073975 (NIH); U01DK073985 (NIH); U01DK074007 (NIH); U01DK073974 (NIH); U01DK074008 (NIH); U01DK074035 (NIH)
Record Dates: First submitted 2010-06-22; First posted 2010-06-23 (Estimated); Results first posted 2019-05-08 (Actual); Last update posted 2019-05-08 (Actual); Status verified 2017-03

CONDITIONS: Gastroparesis
Keywords: gastroparesis; nausea; vomiting
MeSH Terms: conditions — Gastroparesis; Nausea; Vomiting | interventions — Aprepitant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aprepitant (Active Comparator): Aprepitant 125 mg per day
  Interventions: Drug: Aprepitant
- Aprepitant-placebo (Placebo Comparator): Placebo aprepitant 125mg per day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aprepitant — Aprepitant, 125 mg, 1 capsule, q.d. (everyday) with lunch for 4 weeks
  Other Names: Emend
  Arms: Aprepitant
Drug: Placebo — Aprepitant-placebo, 125 mg, 1 capsule, q.d. (everyday) with lunch for 4 weeks
  Arms: Aprepitant-placebo

SUMMARY:
The principal objective of this multicenter, randomized, placebo-controlled trial is to evaluate whether 4 weeks of treatment with aprepitant will improve nausea as compared with placebo in patients with symptoms of chronic nausea and vomiting of presumed gastric origin.

DETAILED DESCRIPTION:
APRON is a multicenter, randomized, double-masked, placebo controlled trial of 4 weeks of treatment with aprepitant or placebo for patients with symptoms of gastroparesis and related disorders. Screening for eligibility and collection of baseline data will span up to 4 weeks after obtaining informed consent and registration. Eligible patients will consist of patients with symptoms of gastroparesis and will be randomized to either aprepitant (125 mg per day) or placebo for 4 weeks.

The symptoms will be measured with the Gastroparesis Cardinal Symptom Index Daily Diary (GCSIDD) for one week at baseline and for four weeks after randomization. In addition, the nausea symptom will be measured daily on a 0 to 100 mm visual analog scale (VAS) for one week at baseline and daily for four weeks after randomization. There will be a 2 week washout period at the end of the treatment to ensure patient safety following the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older at registration
* Gastric emptying scintigraphy within 2 years of registration
* Normal upper endoscopy or upper GI series within 2 years of registration
* Symptoms of chronic nausea or vomiting compatible with gastroparesis or other functional gastric disorder for at least 6 months (does not have to be contiguous) prior to registration with Gastroparesis Cardinal Symptom Index (GCSI) score of greater than or equal to 21
* Significant nausea defined with a visual analog scale (VAS) score of greater than or equal to 25 mm on a 0 to 100 mm scale

Exclusion Criteria:

* Another active disorder which could explain symptoms in the opinion of the investigator
* Use of narcotics more than 3 days per week
* Significant hepatic injury as defined by significant alanine aminotransferase (ALT) and aspartate aminotransferase (AST) elevations of greater than 2x the upper limit of normal (ULN) or a Child-Pugh score of 10 or greater
* Contraindications to aprepitant such as hypersensitivity or allergy
* Concurrent use of warfarin, pimozide, terfenadine, astemizole, or cisapride
* Pregnancy or nursing
* Any other condition, which in the opinion of the investigator would impede compliance or hinder the completion of the study
* Failure to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2013-04; Primary Completion 2015-08 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank Hamilton, MD, MPH, Study Director — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (8):
- United States (8):
  - California Pacific Medical Center, San Francisco, California
  - Stanford University, Stanford, California
  - University of Louisville, Louisville, Kentucky
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Texas Tech University Health Sciences Center, El Paso, Texas

IPD SHARING:
Plan to Share IPD: Yes
Data will be deposited with the NIDDK Data Repository at the end of the funding cycle.
Supporting Information: Study Protocol, CSR, Analytic Code
Time Frame: The primary analysis analytic dataset will be available at the NIDDK Central Repository approximately 6 months after publication. The complete study dataset is due approximately 2 years post study publication.
Access Criteria: The NIDDDK Central Repository staff is responsible for review of requests for use of the APRON public access datasets. A NIDDK SDUC form must be submitted.
URL: https://www.niddkrepository.org/home/

REFERENCES:
- [Derived] Pasricha PJ, Yates KP, Sarosiek I, McCallum RW, Abell TL, Koch KL, Nguyen LAB, Snape WJ, Hasler WL, Clarke JO, Dhalla S, Stein EM, Lee LA, Miriel LA, Van Natta ML, Grover M, Farrugia G, Tonascia J, Hamilton FA, Parkman HP; NIDDK Gastroparesis Clinical Research Consortium (GpCRC). Aprepitant Has Mixed Effects on Nausea and Reduces Other Symptoms in Patients With Gastroparesis and Related Disorders. Gastroenterology. 2018 Jan;154(1):65-76.e11. doi: 10.1053/j.gastro.2017.08.033. Epub 2017 Oct 28. PMID 29111115
- See also: Gastroparesis Clinical Research Consortium website — https://jhuccs1.us/gpcrc/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between April 2013 and July 2015, 126 patients were enrolled at eight participating medical centers, of whom 63 were randomized to aprepitant and 63 to placebo
Pre-assignment Details: Adults, 18 years or older, with symptoms compatible with gastroparesis for 6 months, who had a 4-hour gastric emptying scintigraphy test and a total score >21 on the Gastroparesis Cardinal Symptom Index (GCSI) and a visual analog scale (VAS) mean score of nausea after 7 days of >25 mm on a 0 to 100 mm scale were considered for enrollment.
Period: Overall Study
Arm/Group | Aprepitant | Aprepitant-placebo
Started | 63 | 63
Completed | 57 | 60
Not Completed | 6 | 3
Not completed — Adverse Event | 6 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aprepitant | Aprepitant-placebo | Total
Number analyzed (Participants) | 63 | 63 | 126
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.9 (14.8) | 46.8 (13.5) | 44.8 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 52 | 101
  Male | 14 | 11 | 25
Race/Ethnicity, Customized [Number; unit: participants]
  White | 53 | 59 | 112
  Black | 8 | 2 | 10
  Other | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 63 | 63 | 126
Diabetes type 1 or type 2, No. [Number; unit: participants]
  Have diabetes type 1 or type 2 | 24 | 13 | 37
  Do not have diabetes type 1 or type 2 | 39 | 50 | 89
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 27.8 (8.3) | 28.0 (7.5) | 27.9 (7.9)
Weight [Mean (Standard Deviation); unit: kg] | 75.4 (22.8) | 75.1 (20.6) | 75.2 (21.7)
Waist circumference [Mean (Standard Deviation); unit: cm] | 90.9 (17.2) | 91.3 (18.0) | 91.1 (17.5)
Waist to hip ratio [Mean (Standard Deviation); unit: ratio] | 0.9 (0.1) | 0.9 (0.1) | 0.9 (0.1)
Systolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 121.1 (17.8) | 122.1 (15.0) | 121.6 (16.4)
Diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 73.6 (11.6) | 75.0 (11.3) | 74.3 (11.4)
Medications in past month: proton pump inhibitors [Number; unit: participants]
  Took medication | 42 | 51 | 93
  Did not take medication | 21 | 12 | 33
Medications in past month: benzodiazepine or anxiolytic [Number; unit: participants]
  Took medication | 13 | 27 | 40
  Did not take medication | 50 | 36 | 86
Medications in past month: prokinetic [Number; unit: participants]
  Took medication | 25 | 18 | 43
  Did not take medication | 38 | 45 | 83
Medications in past month: antiemetic [Number; unit: participants]
  Took medication | 44 | 49 | 93
  Did not take medication | 19 | 14 | 33
Medications in past month: selective serotonin reuptake inhibitors (SSRI) [Number; unit: participants]
  Took medication | 9 | 18 | 27
  Did not take medication | 54 | 45 | 99
Medications in past month: tricyclic antidepressant (TCA) [Number; unit: participants]
  Took medication | 11 | 16 | 27
  Did not take medication | 52 | 47 | 99
Medications in past month: other antidepressant [Number; unit: participants]
  Took medication | 12 | 10 | 22
  Did not take medication | 51 | 53 | 104
Medications in past month: narcotic [Number; unit: participants]
  Took medication | 6 | 4 | 10
  Did not take medication | 57 | 59 | 116
Medications in past month: neuropathic or pain modulator... [Number; unit: participants] — Participants who took medications in past month: neuropathic or pain modulator, anti-seizure, or other psychiatric medication
  participants
    Took medication | 27 | 29 | 56
    Did not take medication | 36 | 34 | 70
7-day nausea visual analog scale (VAS) score [Mean (Standard Deviation); unit: units on a scale] — The 7-Day Nausea Visual Analog Scale (VAS) measures severity of current nausea, ranging from a minimum value of 0 (no nausea) to a maximum value of 100 (severe nausea). Higher scores are considered a worse outcome. The VAS is a line measuring 100mm in length. For 7 consecutive days, participants mark their severity of nausea with a vertical line at the point they feel represents their current severity of nausea. The distance to the vertical line is measured with a ruler to the nearest millimeter. The values presented are the mean of the 7 measurements.
  units on a scale | 63.0 (21.5) | 64.1 (20.2) | 63.6 (20.8)
Gastroparesis Cardinal Symptom Index Daily Diary (GCSI-DD): Nausea [Mean (Standard Deviation); unit: hours of nausea] — Gastroparesis Cardinal Symptom Index Daily Diary (GCSI-DD): Nausea is the participant's assessment of the number of hours of nausea experienced in the past 24 hours. The range is 0 to 24 hours.
  hours of nausea | 9.0 (7.0) | 9.3 (7.1) | 9.2 (7.1)
Gastroparesis Cardinal Symptom Index Daily Diary (GCSI-DD): GCSI total score [Mean (Standard Deviation); unit: units on a scale] — The Gastroparesis Cardinal Symptom Index Daily Diary (GCSI-DD): GCSI total score is the average of 3 subscores: Nausea (average of two items: nausea and vomiting), Early Satiety (average of two items: not able to finish normal size meal and feeling excessively full after meals), and Bloating (feeling like you need to loosen your clothes). Each item is the participant's assessment of severity of the symptom during the past 24 hours, where 0=none, 1=mild, 2=moderate, 3=severe, and 4=very severe. The range of scores is 0 to 4, where higher scores are considered a worse outcome.
  units on a scale | 2.2 (0.9) | 2.3 (0.7) | 2.3 (0.8)
Gastroparesis Cardinal Symptom Index Daily Diary (GCSI-DD): Nausea severity [Mean (Standard Deviation); unit: units on a scale] — Gastroparesis Cardinal Symptom Index Daily Diary (GCSI-DD): Nausea severity is the participant's assessment of nausea (feeling sick to your stomach as if you were going to vomit or throw up) during the past 24 hours, where 0=none, 1=mild, 2=moderate, 3=severe, and 4=very severe. The range of scores is 0 to 4, where higher scores are considered a worse outcome.
  units on a scale | 2.6 (0.8) | 2.6 (0.8) | 2.6 (0.8)
Gastroparesis Cardinal Symptom Index Daily Diary (GCSI-DD): Vomiting severity [Mean (Standard Deviation); unit: units on a scale] — Gastroparesis Cardinal Symptom Index Daily Diary (GCSI-DD): Vomiting severity is the participant's assessment of vomiting during the past 24 hours, where 0=none, 1=mild, 2=moderate, 3=severe, and 4=very severe. The range of scores is 0 to 4, where higher scores are considered a worse outcome.
  units on a scale | 1.0 (1.0) | 0.9 (1.0) | 1.0 (1.0)
Gastroparesis Cardinal Symptom Index Daily Diary (GCSI-DD): Early satiety severity [Mean (Standard Deviation); unit: units on a scale] — Gastroparesis Cardinal Symptom Index Daily Diary (GCSI-DD): Early Satiety is the participant's assessment of early satiety (not able to finish a normal-size meal) during the past 24 hours, where 0=none, 1=mild, 2=moderate, 3=severe, and 4=very severe. The range of scores is 0 to 4, where higher scores are considered a worse outcome.
  units on a scale | 2.6 (1.1) | 2.7 (0.9) | 2.6 (1.0)
Gastroparesis Cardinal Symptom Index Daily Diary (GCSI-DD): Excessive fullness severity [Mean (Standard Deviation); unit: units on a scale] — Gastroparesis Cardinal Symptom Index Daily Diary (GCSI-DD): Excessive fullness is the participant's assessment of fullness (feel excessively full after meals) during the past 24 hours, where 0=none, 1=mild, 2=moderate, 3=severe, and 4=very severe. The range of scores is 0 to 4, where higher scores are considered a worse outcome.
  units on a scale | 2.7 (1.1) | 2.8 (0.9) | 2.7 (1.0)
Gastroparesis Cardinal Symptom Index Daily Diary (GCSI-DD): Bloating severity [Mean (Standard Deviation); unit: units on a scale] — Gastroparesis Cardinal Symptom Index Daily Diary (GCSI-DD): Bloating is the participant's assessment of bloating (feeling like you need to loosen your clothes) during the past 24 hours, where 0=none, 1=mild, 2=moderate, 3=severe, and 4=very severe. The range of scores is 0 to 4, where higher scores are considered a worse outcome.
  units on a scale | 2.2 (1.4) | 2.6 (1.1) | 2.4 (1.2)
Gastroparesis Cardinal Symptom Index Daily Diary (GCSI-DD): Upper abdominal pain severity [Mean (Standard Deviation); unit: units on a scale] — Gastroparesis Cardinal Symptom Index Daily Diary (GCSI-DD): Upper abdominal pain is the participant's assessment of upper abdominal pain (above the navel) during the past 24 hours, where 0=none, 1=mild, 2=moderate, 3=severe, and 4=very severe. The range of scores is 0 to 4, where higher scores are considered a worse outcome.
  units on a scale | 2.3 (1.2) | 2.3 (1.0) | 2.3 (1.1)
Gastroparesis Cardinal Symptom Index Daily Diary (GCSI-DD): Vomiting (No. episodes) [Mean (Standard Deviation); unit: number of episodes] — Gastroparesis Cardinal Symptom Index Daily Diary (GCSI-DD): Vomiting is the participant's assessment of the number of episodes of vomiting experienced in the past 24 hours.
  number of episodes | 1.3 (1.6) | 1.1 (1.5) | 1.2 (1.5)
Gastroparesis Cardinal Symptom Index Daily Diary (GCSI-DD): Retching (No. episodes) [Mean (Standard Deviation); unit: number of episodes] — Gastroparesis Cardinal Symptom Index Daily Diary (GCSI-DD): Retching is the participant's assessment of the number of episodes of retching (heaving as if to vomit, but nothing comes up) experienced in the past 24 hours.
  number of episodes | 2.0 (2.5) | 2.3 (2.8) | 2.1 (2.6)
Gastroparesis Cardinal Symptom Index Daily Diary (GCSI-DD): Overall symptom severity [Mean (Standard Deviation); unit: units on a scale] — Gastroparesis Cardinal Symptom Index Daily Diary (GCSI-DD): Overall Symptom Severity is the participant's assessment of overall severity of gastroparesis symptoms during the past 24 hours, where 0=none, 1=mild, 2=moderate, 3=severe, and 4=very severe. The range of scores is 0 to 4, where higher scores are considered a worse outcome.
  units on a scale | 2.5 (0.8) | 2.6 (0.7) | 2.6 (0.8)
PAGI-SYM Severity index: Gastroparesis Cardinal Symptom Index (GCSI), total score [Mean (Standard Deviation); unit: units on a scale] — The PAGI-SYM Severity Index: GCSI Total Score is the average of 3 subscores: Nausea (mean of 3 items: nausea, retching, vomiting), Fullness/Early Satiety (mean of 4 items: stomach fullness, not able to finish normal size meal, feeling excessively full after meals, loss of appetite), and Bloating (mean of 2 items: bloating, stomach visibly larger). Each item is the participant's assessment of symptom severity during the past 24 hours, where 0=none, 1=very mild, 2=mild, 3=moderate, 4=severe, and 5=very severe. The range of scores is 0 to 5, where higher scores are considered a worse outcome.
  units on a scale | 3.4 (0.9) | 3.3 (0.7) | 3.4 (0.8)
PAGI-SYM Severity index: Nausea/vomiting severity subscore [Mean (Standard Deviation); unit: units on a scale] — The PAGI-SYM Severity index: Nausea/vomiting severity subscore is the average of 3 items: nausea, retching, and vomiting. Each item is the participant's assessment of severity of the symptom during the past 24 hours, where 0=none, 1=very mild, 2=mild, 3=moderate, 4=severe, and 5=very severe. The range of scores is 0 to 5, where higher scores are considered a worse outcome.
  units on a scale | 3.3 (1.1) | 2.8 (0.9) | 3.0 (1.1)
PAGI-SYM Severity index: Nausea severity [Mean (Standard Deviation); unit: units on a scale] — The PAGI-SYM Severity index: Nausea severity is the participant's assessment of nausea (feeling sick to your stomach as if you were going to vomit or throw up) during the past 24 hours, where 0=none, 1=very mild, 2=mild, 3=moderate, 4=severe, and 5=very severe. The range of scores is 0 to 5, where higher scores are considered a worse outcome.
  units on a scale | 4.2 (0.8) | 4.0 (0.9) | 4.1 (0.9)
PAGI-SYM Severity index: Retching severity [Mean (Standard Deviation); unit: units on a scale] — The PAGI-SYM Severity index: Retching severity is the participant's assessment of retching (heaving as if to vomit, but nothing comes up) during the past 24 hours, where 0=none, 1=very mild, 2=mild, 3=moderate, 4=severe, and 5=very severe. The range of scores is 0 to 5, where higher scores are considered a worse outcome.
  units on a scale | 3.0 (1.6) | 2.6 (1.3) | 2.8 (1.5)
PAGI-SYM Severity index: Vomiting severity [Mean (Standard Deviation); unit: units on a scale] — The PAGI-SYM Severity index: Vomiting severity is the participant's assessment of vomiting during the past 24 hours, where 0=none, 1=very mild, 2=mild, 3=moderate, 4=severe, and 5=very severe. The range of scores is 0 to 5, where higher scores are considered a worse outcome.
  units on a scale | 2.6 (1.8) | 1.9 (1.6) | 2.2 (1.7)
PAGI-SYM Severity index: Fullness/early satiety subscore [Mean (Standard Deviation); unit: units on a scale] — The PAGI-SYM Severity index: Fullness/early satiety subscore is the average of 4 items: stomach fullness, not able to finish normal size meal, felling excessively full after meals, and loss of appetite. Each item is the participant's assessment of severity of the symptom during the past 24 hours, where 0=none, 1=very mild, 2=mild, 3=moderate, 4=severe, and 5=very severe. The range of scores is 0 to 5, where higher scores are considered a worse outcome.
  units on a scale | 3.7 (1.0) | 3.7 (0.8) | 3.7 (0.9)
PAGI-SYM Severity index: Bloating subscore [Mean (Standard Deviation); unit: units on a scale] — The PAGI-SYM Severity index: Bloating subscore is the average of 2 items: bloating (feeling like you need to loosen your clothes) and stomach visibly larger. Each item is the participant's assessment of severity of the symptom during the past 24 hours, where 0=none, 1=very mild, 2=mild, 3=moderate, 4=severe, and 5=very severe. The range of scores is 0 to 5, where higher scores are considered a worse outcome.
  units on a scale | 3.3 (1.4) | 3.4 (1.4) | 3.4 (1.4)
PAGI-SYM Severity index: Upper abdominal pain subscore [Mean (Standard Deviation); unit: units on a scale] — The PAGI-SYM Severity index: Upper abdominal pain severity is the participant's assessment of upper abdominal pain (above the navel) during the past 24 hours, where 0=none, 1=very mild, 2=mild, 3=moderate, 4=severe, and 5=very severe. The range of scores is 0 to 5, where higher scores are considered a worse outcome.
  units on a scale | 3.4 (1.3) | 3.3 (1.3) | 3.4 (1.3)
PAGI-SYM Severity index: Lower abdominal pain [Mean (Standard Deviation); unit: units on a scale] — The PAGI-SYM Severity index: Lower abdominal pain severity is the participant's assessment of lower abdominal pain (below the navel) during the past 24 hours, where 0=none, 1=very mild, 2=mild, 3=moderate, 4=severe, and 5=very severe. The range of scores is 0 to 5, where higher scores are considered a worse outcome.
  units on a scale | 2.4 (1.6) | 2.5 (1.4) | 2.5 (1.5)
PAGI-SYM Severity index: Lower abdominal discomfort [Mean (Standard Deviation); unit: units on a scale] — The PAGI-SYM Severity index: Lower abdominal discomfort is the participant's assessment of lower abdominal discomfort (below the navel) severity during the past 24 hours, where 0=none, 1=very mild, 2=mild, 3=moderate, 4=severe, and 5=very severe. The range of scores is 0 to 5, where higher scores are considered a worse outcome.
  units on a scale | 2.5 (1.6) | 2.6 (1.4) | 2.6 (1.5)
PAGI-SYM Severity index: Gastroesophageal Reflux (GERD) subscore [Mean (Standard Deviation); unit: units on a scale] — PAGI-SYM Severity index: Gastroesophageal Reflux (GERD) subscore is the average of 7 items (heartburn during day, heartburn lying down, chest discomfort day, chest discomfort during sleep, regurgitation during day, regurgitation lying down, bitter taste in mouth). Each item is the participant's assessment of severity of the symptom, where 0=none, 1=very mild, 2=mild, 3=moderate, 4=severe, and 5=very severe. The range of scores is 0 to 5, where higher scores are considered a worse outcome.
  units on a scale | 2.4 (1.4) | 2.3 (1.4) | 2.3 (1.4)
PAGI-SYM Severity index: Constipation severity [Mean (Standard Deviation); unit: units on a scale] — The PAGI-SYM Severity index: Constipation severity is the participant's assessment of constipation severity during the past 24 hours, where 0=none, 1=very mild, 2=mild, 3=moderate, 4=severe, and 5=very severe. The range of scores is 0 to 5, where higher scores are considered a worse outcome.
  units on a scale | 2.9 (1.7) | 2.6 (1.8) | 2.8 (1.8)
PAGI-SYM Severity index: Diarrhea severity [Mean (Standard Deviation); unit: units on a scale] — The PAGI-SYM Severity index: Diarrhea severity is the participant's assessment of diarrhea severity during the past 24 hours, where 0=none, 1=very mild, 2=mild, 3=moderate, 4=severe, and 5=very severe. The range of scores is 0 to 5, where higher scores are considered a worse outcome.
  units on a scale | 1.6 (1.7) | 1.8 (1.7) | 1.7 (1.7)
PAGI-SYM Severity index: Nausea/vomiting predominant symptom, No. [Number; unit: participants]
  Nausea/vomiting predominant symptom | 38 | 39 | 77
  Nausea/vomiting not predominant symptom | 25 | 24 | 49
Clinical Global Patient Impression Score (patient-rated) [Mean (Standard Deviation); unit: units on a scale] — The Clinical Global Patient Impression Score quantifies the overall relief of the patient's symptom, by asking the participant to consider how they felt over the past week in regard to stomach symptoms and overall well-being, and rate relief of symptoms in comparison to how they felt before entering the study. Possible scores are: -3=very considerably worse, -2=considerably worse, -1=somewhat worse, 0=unchanged, 1=somewhat better, 2=considerably better, 3=completely better. The range of scores is -3 to 3, where higher scores are considered a better outcome.
  units on a scale | -0.6 (1.1) | -0.7 (1.1) | -0.6 (1.1)
Brief Pain Inventory: severity score [Mean (Standard Deviation); unit: units on a scale] — The Brief Pain Inventory: Severity Score is the average of four questions in which the participant rates his or her pain: the worse pain in the past 24 hours, the least pain in the past 24 hours, average pain, and pain right now. The range of possible scores is 0 to 10, with higher scores indicating more severe pain. Higher scores are considered a worse outcome.
  units on a scale | 4.7 (2.5) | 4.6 (2.5) | 4.6 (2.5)
Brief Pain Inventory: Interference score [Mean (Standard Deviation); unit: units on a scale] — The Brief Pain Inventory: Interference Score is the average of seven questions in which the participant rates the degree to which his or her pain interferes with daily functions and mood: general activity, mood, walking ability, normal work, relationships, sleep, enjoyment of life. The range of possible scores is 0 to 10, with higher scores indicating more interference caused by pain. Higher scores are considered a worse outcome.
  units on a scale | 4.4 (3.1) | 5.4 (3.0) | 4.9 (3.1)
Beck Depression Inventory (BDI): Total score [Mean (Standard Deviation); unit: units on a scale] — The Beck Depression Inventory (BDI) survey is comprised of 21 multiple choice questions that relate to depression, cognition, and physical well-being and is extensively used to quantify depression in a range of clinical conditions. The BDI total score is the sum of the 21 items, where each item ranges from 0 to 3 (lower scores are less severe, higher scores are more severe). The range for the BDI total score is 0 to 63, where lower scores indicate less depression and higher scores indicate more sever depression. Higher scores are considered a worse outcome.
  units on a scale | 18.0 (11.8) | 18.3 (12.6) | 18.2 (12.1)
Beck Depression Inventory (BDI): Severe depression, No. [Number; unit: participants] — Severe depression defined as a Beck Depression Inventory (BDI) total score greater than 28 (based on a range of possible scores from 0-63, where higher scores indicate more severe depression).
  participants
    Have severe depression | 11 | 10 | 21
    Do not have severe depression | 52 | 53 | 105
State-Trait Anxiety Inventory (STAI): State anxiety score [Mean (Standard Deviation); unit: units on a scale] — The State-Trait Anxiety Inventory (STAI): State anxiety score is the sum of scores from 20 questions relating to state anxiety, which is a temporary state varying in intensity. The possible range of scores is from 20 to 80, with increasing scores considered a worse outcome.
  units on a scale | 39.6 (13.9) | 41.9 (13.9) | 40.7 (13.9)
State-Trait Anxiety Inventory (STAI): Severe state anxiety, No. [Number; unit: participants]
  Have severe state anxiety | 15 | 19 | 34
  Do not have severe state anxiety | 48 | 44 | 92
State-Trait Anxiety Inventory (STAI): Trait anxiety score [Mean (Standard Deviation); unit: units on a scale] — The State-Trait Anxiety Inventory (STAI): Trait anxiety score is the sum of scores from 20 questions pertaining to trait anxiety, which is a general propensity to be anxious. The possible range of scores is from 20 to 80, with increasing scores considered a worse outcome.
  units on a scale | 40.3 (14.2) | 43.0 (13.2) | 41.6 (13.7)
State-Trait Anxiety Inventory: Severe trait anxiety, No. [Number; unit: participants]
  Have severe trait anxiety | 17 | 19 | 36
  Do not have severe trait anxiety | 46 | 44 | 90
SF-36 Quality of Life (QOL): Physical component summary score [Mean (Standard Deviation); unit: units on a scale] — The SF-36 Quality of Life (QOL) Physical component summary score is the sum of four physical subscores (physical functioning, role-physical, bodily pain, and general health), and is a more general measure of functional health. The range of possible scores is 0 to 100, normalized based on 1998 US population, with higher scores corresponding to higher quality of life.
  units on a scale | 33.5 (9.5) | 29.8 (8.8) | 31.6 (9.4)
SF-36 Quality of Life (QOL): Mental component summary score [Mean (Standard Deviation); unit: units on a scale] — The SF-36 Quality of Life (QOL) Mental component summary score is the sum of four mental subscores (vitality, social functioning, role-emotional, and mental health), and is a more general measure of well-being. The range of possible scores is 0 to 100, normalized based on 1998 US population, with higher scores corresponding to higher quality of life.
  units on a scale | 41.4 (14.3) | 40.5 (13.5) | 40.9 (13.9)
Scintigraphic gastric emptying (GES): Percent gastric retention at 1 hour [Mean (Standard Deviation); unit: percent retention] — Scintigraphic gastric emptying (GES): Percent gastric retention at 1 hour is the percent retention 1 hour after the participant ingests the test meal. The GES is a test performed during screening (baseline) to meet eligibility requirements.
  percent retention | 69.7 (20.0) | 73.0 (19.3) | 71.3 (19.6)
Scintigraphic gastric emptying (GES): Percent gastric retention at 2 hours [Mean (Standard Deviation); unit: percent retention] — Scintigraphic gastric emptying (GES): Percent gastric retention at 2 hours is the percent retention 2 hours after the participant ingests the test meal. The GES is a test performed during screening (baseline) to meet eligibility requirements.
  percent retention | 45.6 (24.9) | 53.1 (23.4) | 49.4 (24.4)
Scintigraphic gastric emptying (GES): Percent gastric retention at 4 hours [Mean (Standard Deviation); unit: percent retention] — Scintigraphic gastric emptying (GES): Percent gastric retention at 4 hours is the percent retention 4 hours after the participant ingests the test meal. The GES is a test performed during screening (baseline) to meet eligibility requirements.
  percent retention | 17.8 (21.8) | 20.4 (17.5) | 19.1 (19.7)
Scintigraphic gastric emptying (GES): Delayed gastric emptying, No. [Number; unit: participants] — Scintigraphic gastric emptying (GES): Delayed gastric emptying is defined as >60% retention 2 hours after the participant ingests the test meal, or >10% retention 4 hours after the participant ingests the test meal.
  participants
    Have delayed gastric emptying | 29 | 43 | 72
    Do not have delayed gastric emptying | 34 | 20 | 54
Scintigraphic gastric emptying (GES): Rapid gastric emptying, No. [Number; unit: participants] — Scintigraphic gastric emptying (GES): Rapid gastric emptying is defined as <30% gastric retention 1 hour after the participant ingests the test meal.
  participants
    Have rapid gastric emptying | 4 | 2 | 6
    Do not have rapid gastric emptying | 59 | 61 | 120

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Improvement in Nausea
Description: The primary outcome measure is a binary (0,1) variable indicating improvement in nausea or not in the mean of available visual analog scale (VAS) scores over the 28 day treatment period compared to the mean of VAS scores during the 7 day baseline period. The criteria for improvement are either a 25 mm or more reduction in mean VAS or attaining a mean VAS during the treatment period of < 25 mm.
Time Frame: 4 weeks
Measure: Number; unit: participants
Arm/Group | Aprepitant | Aprepitant-placebo
Number analyzed (Participants) | 63 | 63
participants | 29 | 25
Statistical Analysis 1: Comparison: Aprepitant vs Aprepitant-placebo; Either 1) improvement in mean of available nausea VAS scores over 28-day treatment period compared to means of VAS during the 7-day baseline (BL) period being ≤ -25 mm, or 2) mean VAS after 28-days of treatment was < 25 mm; Test type: Non-Inferiority or Equivalence — P-values, relative risk ratios, and 95% confidence limits (CI) for the primary ITT were calculated using the Cochran-Mantel-Haenszel chi-square test, stratified by clinic; p = 0.43, Cochran-Mantel-Haenszel; Stratified by clinic; Risk Ratio (RR) = 1.2, 95% CI 2-sided [0.8 to 1.7]

2. Secondary Outcome: Gastroparesis Cardinal Symptom Index Daily Diary (GCSI-DD): Nausea (Hours)
Description: Measure Description: Gastroparesis Cardinal Symptom Index Daily Diary (GCSI-DD): Nausea is the participant's assessment of the number of hours of nausea experienced in the past 24 hours. The range is 0 to 24 hours. The outcome measure, change from baseline in number of hours of nausea, has a possible range from -24 to +24, with negative values indicating a better outcome (improvement) and positive values indicating a worse outcome.
Time Frame: 4 weeks
Population: The smaller number of participants analyzed is due to missing data at the 4-week follow-up visit.
Measure: Mean (Standard Deviation); unit: hours of nausea
Arm/Group | Aprepitant | Aprepitant-placebo
Number analyzed (Participants) | 59 | 63
hours of nausea | -2.5 (3.2) | -1.2 (4.3)
Statistical Analysis 1: Comparison: Aprepitant vs Aprepitant-placebo; Test type: Non-Inferiority or Equivalence — Mean adjusted change from baseline, 95% confidence limits (CI), and P-values were calculated using ANCOVA, regressing change from baseline to 28 days on treatment group and baseline value of the secondary outcome; p = 0.03, ANCOVA; Mean Difference (Net) = -1.5, 95% CI 2-sided [-2.8 to -0.1]

3. Secondary Outcome: Gastroparesis Cardinal Symptom Index Daily Diary (GCSI-DD): Vomiting (No. Episodes)
Description: Gastroparesis Cardinal Symptom Index Daily Diary (GCSI-DD): Vomiting is the participant's assessment of the number of episodes of vomiting experienced in the past 24 hours. The outcome is the change from baseleine in number of times vomited, where negative numbers indicate improvement in vomiting frequency, and positive numbers indicate worsening in vomiting frequency.
Time Frame: 4 weeks
Population: The smaller number of participants analyzed is due to missing data at the 4-week follow-up visit.
Measure: Mean (Standard Deviation); unit: number of episodes
Arm/Group | Aprepitant | Aprepitant-placebo
Number analyzed (Participants) | 59 | 63
number of episodes | -0.5 (1.0) | -0.4 (1.1)
Statistical Analysis 1: Comparison: Aprepitant vs Aprepitant-placebo; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.94, ANCOVA; Mean Difference (Net) = -0.01, 95% CI 2-sided [-0.3 to 0.3]

4. Secondary Outcome: Gastroparesis Cardinal Symptom Index Daily Diary (GCSI-DD): Retching (No. Episodes)
Description: Gastroparesis Cardinal Symptom Index Daily Diary (GCSI-DD): Retching is the participant's assessment of the number of episodes of retching (heaving as if to vomit, but nothing comes up) experienced in the past 24 hours. The outcome is the change from baseline in the number of retching episodes, where negative numbers indicate improvement in retching frequency, and positive numbers indicate worsening in retching frequency.
Time Frame: 4 weeks
Population: The smaller number of participants analyzed is due to missing data at the 4-week follow-up visit.
Measure: Mean (Standard Deviation); unit: number of episodes
Arm/Group | Aprepitant | Aprepitant-placebo
Number analyzed (Participants) | 59 | 63
number of episodes | -0.5 (1.5) | -0.7 (2.0)
Statistical Analysis 1: Comparison: Aprepitant vs Aprepitant-placebo; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.73, ANCOVA; Mean Difference (Net) = 0.1, 95% CI 2-sided [-0.4 to 0.6]

5. Secondary Outcome: Gastroparesis Cardinal Symptom Index Daily Diary (GCSI-DD): GCSI Total Score
Description: The Gastroparesis Cardinal Symptom Index Daily Diary (GCSI-DD): GCSI total score is the average of 3 subscores: Nausea (average of two items: nausea and vomiting), Early Satiety (average of two items: not able to finish normal size meal and feeling excessively full after meals), and Bloating (feeling like you need to loosen your clothes). Each item is the participant's assessment of severity of the symptom during the past 24 hours, where 0=none, 1=mild, 2=moderate, 3=severe, and 4=very severe. The range of scores is 0 to 4, where higher scores are considered a worse outcome. The outcome measure, change from baseline in GCSI total score, has a possible range from -4 to +4, with negative values indicating a better outcome (improvement) and positive values indicating a worse outcome.
Time Frame: 4 weeks
Population: The smaller number of participants analyzed is due to missing data at the 4-week follow-up visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aprepitant | Aprepitant-placebo
Number analyzed (Participants) | 59 | 63
units on a scale | -0.5 (0.9) | -0.4 (0.5)
Statistical Analysis 1: Comparison: Aprepitant vs Aprepitant-placebo; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.22, ANCOVA; Mean Difference (Net) = -0.2, 95% CI 2-sided [-0.4 to 0.1]

6. Secondary Outcome: Gastroparesis Cardinal Symptom Index Daily Diary (GCSI-DD): Nausea Severity
Description: Gastroparesis Cardinal Symptom Index Daily Diary (GCSI-DD): Nausea severity is the participant's assessment of nausea (feeling sick to your stomach as if you were going to vomit or throw up) during the past 24 hours, where 0=none, 1=mild, 2=moderate, 3=severe, and 4=very severe. The range of scores is 0 to 4, where higher scores are considered a worse outcome. The outcome measure, change from baseline in GCSI score, has a possible range from -4 to +4, with negative values indicating a better outcome (improvement) and positive values indicating a worse outcome.
Time Frame: 4 weeks
Population: The smaller number of participants analyzed is due to missing data at the 4-week follow-up visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aprepitant | Aprepitant-placebo
Number analyzed (Participants) | 59 | 63
units on a scale | -0.8 (1.0) | -0.5 (0.7)
Statistical Analysis 1: Comparison: Aprepitant vs Aprepitant-placebo; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.06, ANCOVA; Mean Difference (Net) = -0.3, 95% CI 2-sided [-0.6 to 0.0]

7. Secondary Outcome: Gastroparesis Cardinal Symptom Index Daily Diary (GCSI-DD): Vomiting Severity
Description: Gastroparesis Cardinal Symptom Index Daily Diary (GCSI-DD): Vomiting Severity is the participant's assessment of vomiting during the past 24 hours, where 0=none, 1=mild, 2=moderate, 3=severe, and 4=very severe. The range of scores is 0 to 4, where higher scores are considered a worse outcome. The outcome measure, change from baseline in Vomiting Severity, has a possible range from -4 to +4, with negative values indicating a better outcome (improvement) and positive values indicating a worse outcome.
Time Frame: 4 weeks
Population: The smaller number of participants analyzed is due to missing data at the 4-week follow-up visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aprepitant | Aprepitant-placebo
Number analyzed (Participants) | 59 | 63
units on a scale | -0.4 (0.8) | -0.2 (0.5)
Statistical Analysis 1: Comparison: Aprepitant vs Aprepitant-placebo; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.24, ANCOVA; Mean Difference (Net) = -0.1, 95% CI 2-sided [-0.3 to 0.1]

8. Secondary Outcome: Gastroparesis Cardinal Symptom Index Daily Diary (GCSI-DD): Upper Abdominal Pain Severity
Description: Gastroparesis Cardinal Symptom Index Daily Diary (GCSI-DD): Upper Abdominal Pain Severity is the participant's assessment of upper abdominal pain (above the navel) during the past 24 hours, where 0=none, 1=mild, 2=moderate, 3=severe, and 4=very severe. The range of scores is 0 to 4, where higher scores are considered a worse outcome. The outcome measure, change from baseline in Upper Abdominal Pain Severity, has a possible range from -4 to +4, with negative values indicating a better outcome (improvement) and positive values indicating a worse outcome.
Time Frame: 4 weeks
Population: The smaller number of participants analyzed is due to missing data at the 4-week follow-up visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aprepitant | Aprepitant-placebo
Number analyzed (Participants) | 59 | 63
units on a scale | -0.7 (0.9) | -0.3 (0.7)
Statistical Analysis 1: Comparison: Aprepitant vs Aprepitant-placebo; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.01, ANCOVA; Mean Difference (Net) = -0.4, 95% CI 2-sided [-0.7 to -0.1]

9. Secondary Outcome: Gastroparesis Cardinal Symptom Index Daily Diary (GCSI-DD): Excessive Fullness Severity
Description: Gastroparesis Cardinal Symptom Index Daily Diary (GCSI-DD): Excessive Fullness Severity is the participant's assessment of excessive fullness (feeling excessively full after meals) during the past 24 hours, where 0=none, 1=mild, 2=moderate, 3=severe, and 4=very severe. The range of scores is 0 to 4, where higher scores are considered a worse outcome. The outcome measure, change from baseline in Excessive Fullness Severity, has a possible range from -4 to +4, with negative values indicating a better outcome (improvement) and positive values indicating a worse outcome.
Time Frame: 4 weeks
Population: The smaller number of participants analyzed is due to missing data at the 4-week follow-up visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aprepitant | Aprepitant-placebo
Number analyzed (Participants) | 56 | 61
units on a scale | -0.6 (0.9) | -0.4 (0.7)
Statistical Analysis 1: Comparison: Aprepitant vs Aprepitant-placebo; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.22, ANCOVA; Mean Difference (Net) = -0.2, 95% CI 2-sided [-0.4 to 0.1]

10. Secondary Outcome: Gastroparesis Cardinal Symptom Index Daily Diary (GCSI-DD): Early Satiety Severity
Description: Gastroparesis Cardinal Symptom Index Daily Diary (GCSI-DD): Early Satiety Severity is the participant's assessment of early satiety (not able to finish normal-size meal) during the past 24 hours, where 0=none, 1=mild, 2=moderate, 3=severe, and 4=very severe. The range of scores is 0 to 4, where higher scores are considered a worse outcome. The outcome measure, change from baseline in Early Satiety Severity, has a possible range from -4 to +4, with negative values indicating a better outcome (improvement) and positive values indicating a worse outcome.
Time Frame: 4 weeks
Population: The smaller number of participants analyzed is due to missing data at the 4-week follow-up visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aprepitant | Aprepitant-placebo
Number analyzed (Participants) | 56 | 61
units on a scale | 0.1 (0.2) | 0.08 (0.3)
Statistical Analysis 1: Comparison: Aprepitant vs Aprepitant-placebo; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.51, ANCOVA; Mean Difference (Net) = -0.03, 95% CI 2-sided [-0.1 to 0.1]

11. Secondary Outcome: Gastroparesis Cardinal Symptom Index Daily Diary (GCSI-DD): Bloating Severity
Description: Gastroparesis Cardinal Symptom Index Daily Diary (GCSI-DD): Bloating Severity is the participant's assessment of bloating (feeling like you need to loosen your clothes) during the past 24 hours, where 0=none, 1=mild, 2=moderate, 3=severe, and 4=very severe. The range of scores is 0 to 4, where higher scores are considered a worse outcome. The outcome measure, change from baseline in Bloating Severity, has a possible range from -4 to +4, with negative values indicating a better outcome (improvement) and positive values indicating a worse outcome.
Time Frame: 4 weeks
Population: The smaller number of participants analyzed is due to missing data at the 4-week follow-up visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aprepitant | Aprepitant-placebo
Number analyzed (Participants) | 56 | 61
units on a scale | -0.6 (1.0) | -0.4 (0.8)
Statistical Analysis 1: Comparison: Aprepitant vs Aprepitant-placebo; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.12, ANCOVA; Mean Difference (Net) = -0.2, 95% CI 2-sided [-0.5 to 0.1]

12. Secondary Outcome: Gastroparesis Cardinal Symptom Index Daily Diary (GCSI-DD): Overall Symptom Severity
Description: Gastroparesis Cardinal Symptom Index Daily Diary (GCSI-DD): Overall Symptom Severity is the participant's assessment of overall severity of gastroparesis symptoms during the past 24 hours, where 0=none, 1=mild, 2=moderate, 3=severe, and 4=very severe. The range of scores is 0 to 4, where higher scores are considered a worse outcome. The outcome, change from baseline in Overall Symptom Severity score, has a possible range from -4 to +4, with negative values indicating a better outcome (improvement) and positive values indicating a worse outcome.
Time Frame: 4 weeks
Population: The smaller number of participants analyzed is due to missing data at the 4-week follow-up visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aprepitant | Aprepitant-placebo
Number analyzed (Participants) | 59 | 63
units on a scale | -0.7 (0.8) | -0.4 (0.6)
Statistical Analysis 1: Comparison: Aprepitant vs Aprepitant-placebo; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.02, ANCOVA; Mean Difference (Net) = -0.3, 95% CI 2-sided [-0.6 to -0.1]

13. Secondary Outcome: Clinical Global Patient Impression Score (Patient-rated)
Description: The Clinical Global Patient Impression Score quantifies the overall relief of the patient's symptom, by asking the participant to consider how they felt over the past week in regard to stomach symptoms and overall well-being, and rate relief of symptoms in comparison to how they felt before entering the study. Possible scores are: -3=very considerably worse, -2=considerably worse, -1=somewhat worse, 0=unchanged, 1=somewhat better, 2=considerably better, 3=completely better. The range of scores is -3 to 3, where higher scores are considered a better outcome. The outcome measure, change from baseline in Clinical Global Patient Impression Score, has a possible range of -6 to +6, with positive values indicating a better outcome (improvement) and negative values indicating a worse outcome.
Time Frame: 4 weeks
Population: The smaller number of participants analyzed is due to missing data at the 4-week follow-up visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aprepitant | Aprepitant-placebo
Number analyzed (Participants) | 56 | 61
units on a scale | 1.3 (1.4) | 1.0 (1.4)
Statistical Analysis 1: Comparison: Aprepitant vs Aprepitant-placebo; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.17, ANCOVA; Mean Difference (Net) = 0.3, 95% CI 2-sided [-0.1 to 0.7]

14. Secondary Outcome: Liver Enzymes and Proteins: Alanine Aminotransferase (ALT)
Description: Change from baseline in serum alanine aminotransferase (ALT), U/L
Time Frame: 4 weeks
Population: The smaller number of participants analyzed is due to missing data at the 4-week follow-up visit.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Aprepitant | Aprepitant-placebo
Number analyzed (Participants) | 56 | 61
U/L | 2.3 (36.6) | 0.8 (7.6)
Statistical Analysis 1: Comparison: Aprepitant vs Aprepitant-placebo; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.59, ANCOVA; Mean Difference (Net) = 2.6, 95% CI 2-sided [-7.0 to 12.2]

15. Secondary Outcome: Liver Enzymes and Proteins: Aspartate Aminotransferase (AST)
Description: Change from baseline in aspartate aminotransferase (AST), U/L
Time Frame: 4 weeks
Population: The smaller number of participants analyzed is due to missing data at the 4-week follow-up visit.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Aprepitant | Aprepitant-placebo
Number analyzed (Participants) | 56 | 61
U/L | 3.1 (30.2) | 0.9 (7.7)
Statistical Analysis 1: Comparison: Aprepitant vs Aprepitant-placebo; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.61, ANCOVA; Mean Difference (Net) = 2.1, 95% CI 2-sided [-5.9 to 10.0]

16. Secondary Outcome: Liver Enzymes and Proteins: Total Protein
Description: Change from baseline in total protein (g/dL)
Time Frame: 4 weeks
Population: The smaller number of participants analyzed is due to missing data at the 4-week follow-up visit.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Aprepitant | Aprepitant-placebo
Number analyzed (Participants) | 56 | 61
g/dL | 0.0 (0.4) | -0.1 (0.4)
Statistical Analysis 1: Comparison: Aprepitant vs Aprepitant-placebo; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.23, ANCOVA; Mean Difference (Net) = 0.1, 95% CI 2-sided [-0.1 to 0.2]

17. Secondary Outcome: Hemoglobin A1c (HbA1c)
Description: Change from baseline in hemoglobin A1c (HbA1c) (%)
Time Frame: 4 weeks
Population: The smaller number of participants analyzed is due to missing data at the 4-week follow-up visit.
Measure: Mean (Standard Deviation); unit: percent glycosylated hemoglobin
Arm/Group | Aprepitant | Aprepitant-placebo
Number analyzed (Participants) | 56 | 61
percent glycosylated hemoglobin | -0.1 (1.0) | 0.1 (0.5)
Statistical Analysis 1: Comparison: Aprepitant vs Aprepitant-placebo; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.97, ANCOVA; Mean Difference (Net) = 0.0, 95% CI 2-sided [-0.5 to 0.5]

18. Secondary Outcome: Glucose
Description: Change from baseline in glucose (mg/dL)
Time Frame: 4 weeks
Population: The smaller number of participants analyzed is due to missing data at the 4-week follow-up visit.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Aprepitant | Aprepitant-placebo
Number analyzed (Participants) | 56 | 61
mg/dL | 9.6 (66.8) | 7.0 (44.8)
Statistical Analysis 1: Comparison: Aprepitant vs Aprepitant-placebo; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.77, ANCOVA; Mean Difference (Net) = 3.1, 95% CI 2-sided [-18.0 to 24.2]

19. Secondary Outcome: Liver Enzymes and Proteins: Albumin
Description: Change from baseline in albumin (g/dL)
Time Frame: 4 weeks
Population: The smaller number of participants analyzed is due to missing data at the 4-week follow-up visit.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Aprepitant | Aprepitant-placebo
Number analyzed (Participants) | 56 | 61
g/dL | -0.1 (0.4) | -0.1 (0.4)
Statistical Analysis 1: Comparison: Aprepitant vs Aprepitant-placebo; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.46, ANCOVA; Mean Difference (Net) = -0.1, 95% CI 2-sided [-0.2 to 0.1]

20. Secondary Outcome: Hemoglobin
Description: Change from baseline in hemoglobin (g/dL)
Time Frame: 4 weeks
Population: The smaller number of participants analyzed is due to missing data at the 4-week follow-up visit.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Aprepitant | Aprepitant-placebo
Number analyzed (Participants) | 56 | 61
g/dL | -0.1 (0.9) | -0.2 (0.6)
Statistical Analysis 1: Comparison: Aprepitant vs Aprepitant-placebo; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.44, ANCOVA; Mean Difference (Net) = 0.1, 95% CI 2-sided [-0.2 to 0.4]

21. Secondary Outcome: Hematocrit
Description: Change from baseline in hematocrit
Time Frame: 4 weeks
Population: The smaller number of participants analyzed is due to missing data at the 4-week follow-up visit.
Measure: Mean (Standard Deviation); unit: percentage RBCs
Arm/Group | Aprepitant | Aprepitant-placebo
Number analyzed (Participants) | 56 | 61
percentage RBCs | -0.4 (2.7) | -0.4 (1.9)
Statistical Analysis 1: Comparison: Aprepitant vs Aprepitant-placebo; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.77, ANCOVA; Mean Difference (Net) = 0.1, 95% CI 2-sided [-0.7 to 0.9]

22. Secondary Outcome: White Blood Cell Count (WBC)
Description: Change from baseline in white blood cell count (WBC)
Time Frame: 4 weeks
Population: The smaller number of participants analyzed is due to missing data at the 4-week follow-up visit.
Measure: Mean (Standard Deviation); unit: x10^9 cells/L
Arm/Group | Aprepitant | Aprepitant-placebo
Number analyzed (Participants) | 56 | 61
x10^9 cells/L | -0.3 (1.5) | -0.3 (1.8)
Statistical Analysis 1: Comparison: Aprepitant vs Aprepitant-placebo; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.80, ANCOVA; Mean Difference (Net) = -0.1, 95% CI 2-sided [-0.6 to 0.5]

23. Secondary Outcome: Red Blood Cell Count (RBC)
Description: Change from baseline in red blood cell count (RBC)
Time Frame: 4 weeks
Population: The smaller number of participants analyzed is due to missing data at the 4-week follow-up visit.
Measure: Mean (Standard Deviation); unit: x10^6 cells/microliter
Arm/Group | Aprepitant | Aprepitant-placebo
Number analyzed (Participants) | 56 | 61
x10^6 cells/microliter | -0.1 (0.3) | -0.1 (0.2)
Statistical Analysis 1: Comparison: Aprepitant vs Aprepitant-placebo; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.88, ANCOVA; Mean Difference (Net) = 0.0, 95% CI 2-sided [-0.1 to 0.1]

24. Secondary Outcome: Platelet Count
Description: Change from baseline in platelet count
Time Frame: 4 weeks
Population: The smaller number of participants analyzed is due to missing data at the 4-week follow-up visit.
Measure: Mean (Standard Deviation); unit: x10^3 cells/microliter
Arm/Group | Aprepitant | Aprepitant-placebo
Number analyzed (Participants) | 56 | 61
x10^3 cells/microliter | -7.3 (47.1) | 4.8 (38.5)
Statistical Analysis 1: Comparison: Aprepitant vs Aprepitant-placebo; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.17, ANCOVA; Mean Difference (Net) = -10.9, 95% CI 2-sided [-26.5 to 4.7]

25. Secondary Outcome: Carbon Dioxide
Description: Change from baseline in carbon dioxide (mEg/L)
Time Frame: 4 weeks
Population: The smaller number of participants analyzed is due to missing data at the 4-week follow-up visit.
Measure: Mean (Standard Deviation); unit: mEq/L
Arm/Group | Aprepitant | Aprepitant-placebo
Number analyzed (Participants) | 56 | 61
mEq/L | -0.4 (2.5) | 0.4 (2.4)
Statistical Analysis 1: Comparison: Aprepitant vs Aprepitant-placebo; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.07, ANCOVA; Mean Difference (Net) = -0.7, 95% CI 2-sided [-1.5 to 0.0]

26. Secondary Outcome: Chloride
Description: Change from baseline in chloride (mEq/L)
Time Frame: 4 weeks
Population: The smaller number of participants analyzed is due to missing data at the 4-week follow-up visit.
Measure: Mean (Standard Deviation); unit: mEq/L
Arm/Group | Aprepitant | Aprepitant-placebo
Number analyzed (Participants) | 56 | 61
mEq/L | 0.6 (3.0) | -0.2 (2.9)
Statistical Analysis 1: Comparison: Aprepitant vs Aprepitant-placebo; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.53, ANCOVA; Mean Difference (Net) = 0.3, 95% CI 2-sided [-0.7 to 1.3]

27. Secondary Outcome: Sodium
Description: Change from baseline in sodium (mEq/L)
Time Frame: 4 weeks
Population: The smaller number of participants analyzed is due to missing data at the 4-week follow-up visit.
Measure: Mean (Standard Deviation); unit: mEq/L
Arm/Group | Aprepitant | Aprepitant-placebo
Number analyzed (Participants) | 56 | 61
mEq/L | -0.3 (2.3) | -0.7 (2.9)
Statistical Analysis 1: Comparison: Aprepitant vs Aprepitant-placebo; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.93, ANCOVA; Mean Difference (Net) = 0.0, 95% CI 2-sided [-0.9 to 1.0]

28. Secondary Outcome: Potassium
Description: Change from baseline in potassium (mEq/L)
Time Frame: 4 weeks
Population: The smaller number of participants analyzed is due to missing data at the 4-week follow-up visit.
Measure: Mean (Standard Deviation); unit: mEq/L
Arm/Group | Aprepitant | Aprepitant-placebo
Number analyzed (Participants) | 56 | 61
mEq/L | 0.1 (0.5) | 0.0 (0.4)
Statistical Analysis 1: Comparison: Aprepitant vs Aprepitant-placebo; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.52, ANCOVA; Mean Difference (Net) = 0.0, 95% CI 2-sided [-1.0 to 0.2]

29. Secondary Outcome: Calcium
Description: Change from baseline in calcium (mg/dL)
Time Frame: 4 weeks
Population: The smaller number of participants analyzed is due to missing data at the 4-week follow-up visit.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Aprepitant | Aprepitant-placebo
Number analyzed (Participants) | 56 | 61
mg/dL | -0.1 (0.4) | -0.1 (0.4)
Statistical Analysis 1: Comparison: Aprepitant vs Aprepitant-placebo; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.76, ANCOVA; Mean Difference (Net) = 0.0, 95% CI 2-sided [-0.1 to 0.1]

30. Secondary Outcome: Blood Urea Nitrogen (BUN)
Description: Change from baseline in blood urea nitrogen (BUN) (mg/dL)
Time Frame: 4 weeks
Population: The smaller number of participants analyzed is due to missing data at the 4-week follow-up visit.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Aprepitant | Aprepitant-placebo
Number analyzed (Participants) | 56 | 61
mg/dL | -0.9 (4.6) | -0.3 (3.3)
Statistical Analysis 1: Comparison: Aprepitant vs Aprepitant-placebo; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.45, ANCOVA; Mean Difference (Net) = -0.5, 95% CI 2-sided [-2.0 to 0.9]

31. Secondary Outcome: Magnesium
Description: Change from baseline in magnesium (mg/dL)
Time Frame: 4 weeks
Population: The smaller number of participants analyzed is due to missing data at the 4-week follow-up visit.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Aprepitant | Aprepitant-placebo
Number analyzed (Participants) | 56 | 61
mg/dL | 0.0 (0.2) | -0.0 (0.2)
Statistical Analysis 1: Comparison: Aprepitant vs Aprepitant-placebo; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.18, ANCOVA; Mean Difference (Net) = 0.0, 95% CI 2-sided [0.0 to 0.1]

32. Secondary Outcome: Creatinine
Description: Change from baseline in creatinine (mg/dL)
Time Frame: 4 weeks
Population: The smaller number of participants analyzed is due to missing data at the 4-week follow-up visit.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Aprepitant | Aprepitant-placebo
Number analyzed (Participants) | 56 | 61
mg/dL | -0.1 (0.2) | 0.0 (0.2)
Statistical Analysis 1: Comparison: Aprepitant vs Aprepitant-placebo; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.008, ANCOVA; Mean Difference (Net) = -0.1, 95% CI 2-sided [-0.2 to -0]

33. Secondary Outcome: PAGI-SYM Severity Index: Gastroparesis Cardinal Symptom Index (GCSI) Score
Description: PAGI-SYM Severity index: Gastroparesis Cardinal Symptom Index (GCSI) score is the average of 3 subscores: Nausea (average of 3 items: nausea, retching, and vomiting), Fullness/Early Satiety (average of 4 items: stomach fullness, not able to finish normal size meal, feeling excessively full after meals, and loss of appetite), and Bloating (average if 2 items: bloating and stomach visibly larger). Each item is the participant's assessment of severity of the symptom during the past 24 hours, where 0=none, 1=very mild, 2=mild, 3=moderate, 4=severe, and 5=very severe. The outcome measure, change from baseline in GCSI score, has a possible range from -5 to +5, with negative values indicating a better outcome (improvement) and positive values indicating a worse outcome.
Time Frame: 4 weeks
Population: The smaller number of participants analyzed is due to missing data at the 4-week follow-up visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aprepitant | Aprepitant-placebo
Number analyzed (Participants) | 59 | 63
units on a scale | -1.3 (1.0) | -0.7 (0.9)
Statistical Analysis 1: Comparison: Aprepitant vs Aprepitant-placebo; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.001, ANCOVA; Mean Difference (Net) = -0.6, 95% CI 2-sided [-0.9 to -0.3]

34. Secondary Outcome: PAGI-SYM Severity Index: Nausea/Vomiting Severity Subscore
Description: The PAGI-SYM Severity index: Nausea/vomiting severity subscore is the average of 3 items: nausea, retching, and vomiting. Each item is the participant's assessment of severity of the symptom during the past 24 hours, where 0=none, 1=very mild, 2=mild, 3=moderate, 4=severe, and 5=very severe. The range of scores is 0 to 5, where higher scores are considered a worse outcome. The outcome measure, change from baseline in Nausea/vomiting severity subscore, has a possible range from -5 to +5, with negative values indicating a better outcome (improvement) and positive values indicating a worse outcome.
Time Frame: 4 weeks
Population: The smaller number of participants analyzed is due to missing data at the 4-week follow-up visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aprepitant | Aprepitant-placebo
Number analyzed (Participants) | 59 | 63
units on a scale | -1.7 (1.3) | -0.7 (1.1)
Statistical Analysis 1: Comparison: Aprepitant vs Aprepitant-placebo; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p < 0.001, ANCOVA; Mean Difference (Net) = -0.8, 95% CI 2-sided [-1.2 to -0.4]

35. Secondary Outcome: PAGI-SYM Severity Index: Fullness/Early Satiety Subscore
Description: The PAGI-SYM Severity index: Fullness/Early Satiety Subscore is the average of 4 items: stomach fullness, not able to finish normal size meal, felling excessively full after meals, and loss of appetite. Each item is the participant's assessment of severity of the symptom during the past 24 hours, where 0=none, 1=very mild, 2=mild, 3=moderate, 4=severe, and 5=very severe. The range of scores is 0 to 5, where higher scores are considered a worse outcome. The outcome measure, change from baseline in Fullness/Early Satiety Subscore, has a possible range from -5 to +5, with negative values indicating a better outcome (improvement) and positive values indicating a worse outcome.
Time Frame: 4 weeks
Population: The smaller number of participants analyzed is due to missing data at the 4-week follow-up visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aprepitant | Aprepitant-placebo
Number analyzed (Participants) | 59 | 63
units on a scale | -1.0 (1.3) | -0.7 (1.0)
Statistical Analysis 1: Comparison: Aprepitant vs Aprepitant-placebo; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.13, ANCOVA; Mean Difference (Net) = -0.3, 95% CI 2-sided [-0.7 to 0.1]

36. Secondary Outcome: PAGI-SYM Severity Index: Bloating Subscore
Description: The PAGI-SYM Severity index: Bloating Subscore is the average of 2 items: bloating (feeling like you need to loosen your clothes) and stomach visibly larger. Each item is the participant's assessment of severity of the symptom during the past 24 hours, where 0=none, 1=very mild, 2=mild, 3=moderate, 4=severe, and 5=very severe. The outcome measure, change from baseline in Bloating Subscore, has a possible range from -5 to +5, with negative values indicating a better outcome (improvement) and positive values indicating a worse outcome.
Time Frame: 4 weeks
Population: The smaller number of participants analyzed is due to missing data at the 4-week follow-up visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aprepitant | Aprepitant-placebo
Number analyzed (Participants) | 59 | 63
units on a scale | -1.2 (1.2) | -0.6 (1.2)
Statistical Analysis 1: Comparison: Aprepitant vs Aprepitant-placebo; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.004, ANCOVA; Mean Difference (Net) = -0.6, 95% CI 2-sided [-1.2 to -0.2]

37. Secondary Outcome: PAGI-SYM Severity Index: Upper Abdominal Pain Subscore
Description: The PAGI-SYM Severity index: Upper Abdominal Pain subscore is the average of 2 items (upper abdominal pain, upper abdominal discomfort). Each item is the participant's assessment of severity of the symptom during the past 24 hours, where 0=none, 1=very mild, 2=mild, 3=moderate, 4=severe, and 5=very severe. The range of scores is 0 to 5, where higher scores are considered a worse outcome. The outcome measure, change from baseline in Upper Abdominal Pain Subscore, has a possible range from -5 to +5, with negative values indicating a better outcome (improvement) and positive values indicating a worse outcome.
Time Frame: 4 weeks
Population: The smaller number of participants analyzed is due to missing data at the 4-week follow-up visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aprepitant | Aprepitant-placebo
Number analyzed (Participants) | 59 | 63
units on a scale | -1.1 (1.5) | -0.6 (1.2)
Statistical Analysis 1: Comparison: Aprepitant vs Aprepitant-placebo; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.08, ANCOVA; Mean Difference (Net) = -0.4, 95% CI 2-sided [-0.9 to 0.1]

38. Secondary Outcome: PAGI-SYM Severity Index: GERD Subscore
Description: PAGI-SYM Severity index: Gastroesophageal Reflux (GERD) Subscore is the average of 7 items (heartburn during day, heartburn lying down, chest discomfort day, chest discomfort during sleep, regurgitation during day, regurgitation lying down, bitter taste in mouth). Each item is the participant's assessment of severity of the symptom, where 0=none, 1=very mild, 2=mild, 3=moderate, 4=severe, and 5=very severe. The range of scores is 0 to 5, where higher scores are considered a worse outcome. The outcome measure, change from baseline in GERD Subscore, has a possible range from -5 to +5, with negative values indicating a better outcome (improvement) and positive values indicating a worse outcome.
Time Frame: 4 weeks
Population: The smaller number of participants analyzed is due to missing data at the 4-week follow-up visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aprepitant | Aprepitant-placebo
Number analyzed (Participants) | 59 | 63
units on a scale | -1.1 (1.3) | -0.6 (0.9)
Statistical Analysis 1: Comparison: Aprepitant vs Aprepitant-placebo; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.007, ANCOVA; Mean Difference (Net) = -0.5, 95% CI 2-sided [-0.8 to -0.1]

39. Secondary Outcome: PAGI-SYM Severity Index: Nausea Severity
Description: The PAGI-SYM Severity index: Nausea severity is the participant's assessment of nausea (feeling sick to your stomach as if you were going to vomit or throw up) during the past 24 hours, where 0=none, 1=very mild, 2=mild, 3=moderate, 4=severe, and 5=very severe. The range of scores is 0 to 5, where higher scores are considered a worse outcome. The outcome measure, change from baseline in Nausea Severity, has a possible range from -5 to +5, with negative values indicating a better outcome (improvement) and positive values indicating a worse outcome.
Time Frame: 4 weeks
Population: The smaller number of participants analyzed is due to missing data at the 4-week follow-up visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aprepitant | Aprepitant-placebo
Number analyzed (Participants) | 59 | 63
units on a scale | -1.8 (1.5) | -1.0 (1.4)
Statistical Analysis 1: Comparison: Aprepitant vs Aprepitant-placebo; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.005, ANCOVA; Mean Difference (Net) = -0.7, 95% CI 2-sided [-1.3 to -0.2]

40. Secondary Outcome: PAGI-SYM Severity Index: Vomiting Severity
Description: The PAGI-SYM Severity index: Vomiting Severity is the participant's assessment of vomiting during the past 24 hours, where 0=none, 1=very mild, 2=mild, 3=moderate, 4=severe, and 5=very severe. The range of scores is 0 to 5, where higher scores are considered a worse outcome. The outcome measure, change from baseline in Vomiting Severity, has a possible range from -5 to +5, with negative values indicating a better outcome (improvement) and positive values indicating a worse outcome.
Time Frame: 4 weeks
Population: The smaller number of participants analyzed is due to missing data at the 4-week follow-up visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aprepitant | Aprepitant-placebo
Number analyzed (Participants) | 59 | 63
units on a scale | -1.6 (1.7) | -0.5 (1.4)
Statistical Analysis 1: Comparison: Aprepitant vs Aprepitant-placebo; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.001, ANCOVA; Mean Difference (Net) = -0.7, 95% CI 2-sided [-1.1 to -0.3]

41. Secondary Outcome: PAGI-SYM Severity Index: Retching Severity
Description: The PAGI-SYM Severity index: Retching Severity is the participant's assessment of retching (heaving as if to vomit, but nothing comes up) during the past 24 hours, where 0=none, 1=very mild, 2=mild, 3=moderate, 4=severe, and 5=very severe. The range of scores is 0 to 5, where higher scores are considered a worse outcome. The outcome measure, change from baseline in Retching Severity, has a possible range from -5 to +5, with negative values indicating a better outcome (improvement) and positive values indicating a worse outcome.
Time Frame: 4 weeks
Population: The smaller number of participants analyzed is due to missing data at the 4-week follow-up visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aprepitant | Aprepitant-placebo
Number analyzed (Participants) | 59 | 63
units on a scale | -1.7 (1.6) | -0.8 (1.4)
Statistical Analysis 1: Comparison: Aprepitant vs Aprepitant-placebo; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.003, ANCOVA; Mean Difference (Net) = -0.8, 95% CI 2-sided [-2.3 to -0.3]

42. Secondary Outcome: PAGI-SYM Severity Index: Stomach Fullness Severity
Description: PAGI-SYM Severity index: Stomach Fullness severity is the participant's assessment of stomach fullness during the past 24 hours, where 0=none, 1=very mild, 2=mild, 3=moderate, 4=severe, and 5=very severe. The range of scores is 0 to 5, where higher scores are considered a worse outcome. The outcome measure, change from baseline in Stomach Fullness severity, has a possible range from -5 to +5, with negative values indicating a better outcome (improvement) and positive values indicating a worse outcome.
Time Frame: 4 weeks
Population: The smaller number of participants analyzed is due to missing data at the 4-week follow-up visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aprepitant | Aprepitant-placebo
Number analyzed (Participants) | 56 | 61
units on a scale | -1.1 (1.6) | -0.5 (1.4)
Statistical Analysis 1: Comparison: Aprepitant vs Aprepitant-placebo; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.03, ANCOVA; Mean Difference (Net) = -0.5, 95% CI 2-sided [-1.0 to -0.1]

43. Secondary Outcome: PAGI-SYM Severity Index: Unable to Finish Meal Severity
Description: PAGI-SYM Severity index: Unable to Finish Meal severity is the participant's assessment of being unable to finish a normal size meal during the past 24 hours, where 0=none, 1=very mild, 2=mild, 3=moderate, 4=severe, and 5=very severe. The range of scores is 0 to 5, where higher scores are considered a worse outcome. The outcome measure, change from baseline in Unable to Finish Meal severity, has a possible range from -5 to +5, with negative values indicating a better outcome (improvement) and positive values indicating a worse outcome.
Time Frame: 4 weeks
Population: The smaller number of participants analyzed is due to missing data at the 4-week follow-up visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aprepitant | Aprepitant-placebo
Number analyzed (Participants) | 56 | 61
units on a scale | -0.8 (1.4) | -0.6 (1.3)
Statistical Analysis 1: Comparison: Aprepitant vs Aprepitant-placebo; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.16, ANCOVA; Mean Difference (Net) = -0.3, 95% CI 2-sided [-0.8 to 0.1]

44. Secondary Outcome: PAGI-SYM Severity Index: Excessive Fullness Severity
Description: PAGI-SYM Severity index: Excessive fullness severity is the participant's assessment of feeling excessively full after meals during the past 24 hours, where 0=none, 1=very mild, 2=mild, 3=moderate, 4=severe, and 5=very severe. The range of scores is 0 to 5, where higher scores are considered a worse outcome. The outcome measure, change from baseline in Excessive Fullness severity, has a possible range from -5 to +5, with negative values indicating a better outcome (improvement) and positive values indicating a worse outcome.
Time Frame: 4 weeks
Population: The smaller number of participants analyzed is due to missing data at the 4-week follow-up visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aprepitant | Aprepitant-placebo
Number analyzed (Participants) | 56 | 61
units on a scale | -1.1 (1.4) | -0.6 (1.2)
Statistical Analysis 1: Comparison: Aprepitant vs Aprepitant-placebo; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.05, ANCOVA; Mean Difference (Net) = -0.5, 95% CI 2-sided [-0.9 to 0.0]

45. Secondary Outcome: PAGI-SYM Severity Index: Loss of Appetite Severity
Description: PAGI-SYM Severity index: Loss of appetite severity is the participant's assessment of loss of appetite during the past 24 hours, where 0=none, 1=very mild, 2=mild, 3=moderate, 4=severe, and 5=very severe. The range of scores is 0 to 5, where higher scores are considered a worse outcome. The outcome measure, change from baseline in Loss of appetite severity, has a possible range from -5 to +5, with negative values indicating a better outcome (improvement) and positive values indicating a worse outcome.
Time Frame: 4 weeks
Population: The smaller number of participants analyzed is due to missing data at the 4-week follow-up visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aprepitant | Aprepitant-placebo
Number analyzed (Participants) | 56 | 61
units on a scale | -0.9 (1.6) | -0.9 (1.4)
Statistical Analysis 1: Comparison: Aprepitant vs Aprepitant-placebo; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.72, ANCOVA; Mean Difference (Net) = 0.1, 95% CI 2-sided [-0.4 to 0.6]

46. Secondary Outcome: PAGI-SYM Severity Index: Bloating Severity
Description: The PAGI-SYM Severity index: Bloating Severity is the participant's assessment of bloating (feel like you need to loosen your clothes) during the past 24 hours, where 0=none, 1=very mild, 2=mild, 3=moderate, 4=severe, and 5=very severe. The range of scores is 0 to 5, where higher scores are considered a worse outcome. The outcome measure, change from baseline in Bloating Severity, has a possible range from -5 to +5, with negative values indicating a better outcome (improvement) and positive values indicating a worse outcome.
Time Frame: 4 weeks
Population: The smaller number of participants analyzed is due to missing data at the 4-week follow-up visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aprepitant | Aprepitant-placebo
Number analyzed (Participants) | 56 | 61
units on a scale | -1.2 (1.4) | -0.5 (1.3)
Statistical Analysis 1: Comparison: Aprepitant vs Aprepitant-placebo; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.001, ANCOVA; Mean Difference (Net) = -0.8, 95% CI 2-sided [-1.2 to -0.3]

47. Secondary Outcome: PAGI-SYM Severity Index: Stomach Distention Severity
Description: The PAGI-SYM Severity index: Stomach distention severity is the participant's assessment of stomach distention (stomach or belly visibly larger) during the past 24 hours, where 0=none, 1=very mild, 2=mild, 3=moderate, 4=severe, and 5=very severe. The range of scores is 0 to 5, where higher scores are considered a worse outcome. The outcome measure, change from baseline in Stomach Distention severity, has a possible range from -5 to +5, with negative values indicating a better outcome (improvement) and positive values indicating a worse outcome.
Time Frame: 4 weeks
Population: The smaller number of participants analyzed is due to missing data at the 4-week follow-up visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aprepitant | Aprepitant-placebo
Number analyzed (Participants) | 56 | 61
units on a scale | -1.1 (1.3) | -0.7 (1.3)
Statistical Analysis 1: Comparison: Aprepitant vs Aprepitant-placebo; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.04, ANCOVA; Mean Difference (Net) = -0.5, 95% CI 2-sided [-0.9 to 0.0]

48. Secondary Outcome: PAGI-SYM Severity Index: Upper Abdominal Pain Severity
Description: The PAGI-SYM Severity index: Upper Abdominal Pain severity is the participant's assessment of upper abdominal pain (above the navel) during the past 24 hours, where 0=none, 1=very mild, 2=mild, 3=moderate, 4=severe, and 5=very severe. The range of scores is 0 to 5, where higher scores are considered a worse outcome. The outcome measure, change from baseline in Upper Abdominal Pain severity, has a possible range from -5 to +5, with negative values indicating a better outcome (improvement) and positive values indicating a worse outcome.
Time Frame: 4 weeks
Population: The smaller number of participants analyzed is due to missing data at the 4-week follow-up visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aprepitant | Aprepitant-placebo
Number analyzed (Participants) | 56 | 61
units on a scale | -1.0 (1.6) | -0.5 (1.4)
Statistical Analysis 1: Comparison: Aprepitant vs Aprepitant-placebo; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.14, ANCOVA; Mean Difference (Net) = -0.4, 95% CI 2-sided [-0.9 to 0.1]

49. Secondary Outcome: PAGI-SYM Severity Index: Upper Abdominal Discomfort Severity
Description: The PAGI-SYM Severity index: Upper Abdominal Discomfort severity is the participant's assessment of upper abdominal discomfort (above the navel) during the past 24 hours, where 0=none, 1=very mild, 2=mild, 3=moderate, 4=severe, and 5=very severe. The range of scores is 0 to 5, where higher scores are considered a worse outcome. The outcome measure, change from baseline in Upper Abdominal Discomfort severity, has a possible range from -5 to +5, with negative values indicating a better outcome (improvement) and positive values indicating a worse outcome.
Time Frame: 4 weeks
Population: The smaller number of participants analyzed is due to missing data at the 4-week follow-up visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aprepitant | Aprepitant-placebo
Number analyzed (Participants) | 56 | 61
units on a scale | -1.2 (1.6) | -0.7 (1.3)
Statistical Analysis 1: Comparison: Aprepitant vs Aprepitant-placebo; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.07, ANCOVA; Mean Difference (Net) = -0.5, 95% CI 2-sided [-1.0 to 0.0]

50. Secondary Outcome: PAGI-SYM Severity Index: Lower Abdominal Pain Severity
Description: The PAGI-SYM Severity index: Lower Abdominal Pain severity is the participant's assessment of lower abdominal pain (below the navel) during the past 24 hours, where 0=none, 1=very mild, 2=mild, 3=moderate, 4=severe, and 5=very severe. The range of scores is 0 to 5, where higher scores are considered a worse outcome. The outcome measure, change from baseline in Lower Abdominal Pain severity, has a possible range from -5 to +5, with negative values indicating a better outcome (improvement) and positive values indicating a worse outcome.
Time Frame: 4 weeks
Population: The smaller number of participants analyzed is due to missing data at the 4-week follow-up visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aprepitant | Aprepitant-placebo
Number analyzed (Participants) | 56 | 61
units on a scale | -0.8 (1.4) | -0.6 (1.5)
Statistical Analysis 1: Comparison: Aprepitant vs Aprepitant-placebo; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.19, ANCOVA; Mean Difference (Net) = -0.3, 95% CI 2-sided [-0.8 to 0.2]

51. Secondary Outcome: PAGI-SYM Severity Index: Lower Abdominal Discomfort Severity
Description: The PAGI-SYM Severity index: Lower Abdominal Discomfort severity is the participant's assessment of lower abdominal discomfort (below the navel) during the past 24 hours, where 0=none, 1=very mild, 2=mild, 3=moderate, 4=severe, and 5=very severe. The range of scores is 0 to 5, where higher scores are considered a worse outcome. The outcome measure, change from baseline in Lower Abdominal Discomfort severity, has a possible range from -5 to +5, with negative values indicating a better outcome (improvement) and positive values indicating a worse outcome.
Time Frame: 4 weeks
Population: The smaller number of participants analyzed is due to missing data at the 4-week follow-up visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aprepitant | Aprepitant-placebo
Number analyzed (Participants) | 56 | 61
units on a scale | -1.1 (1.4) | -0.6 (1.5)
Statistical Analysis 1: Comparison: Aprepitant vs Aprepitant-placebo; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.04, ANCOVA; Mean Difference (Net) = -0.5, 95% CI 2-sided [-0.9 to -0.0]

52. Secondary Outcome: PAGI-SYM Severity Index: Heartburn During the Day Severity
Description: The PAGI-SYM Severity index: Heartburn during the day severity is the participant's assessment of heartburn (burning pain rising in your chest or throat) during the day over the past 24 hours, where 0=none, 1=very mild, 2=mild, 3=moderate, 4=severe, and 5=very severe. The range of scores is 0 to 5, where higher scores are considered a worse outcome. The outcome measure, change from baseline in Heartburn During the Day severity, has a possible range from -5 to +5, with negative values indicating a better outcome (improvement) and positive values indicating a worse outcome.
Time Frame: 4 weeks
Population: The smaller number of participants analyzed is due to missing data at the 4-week follow-up visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aprepitant | Aprepitant-placebo
Number analyzed (Participants) | 56 | 61
units on a scale | -1.2 (1.5) | -0.6 (1.4)
Statistical Analysis 1: Comparison: Aprepitant vs Aprepitant-placebo; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.02, ANCOVA; Mean Difference (Net) = -0.5, 95% CI 2-sided [-1.0 to -0.1]

53. Secondary Outcome: PAGI-SYM Severity Index: Heartburn When Lying Down Severity
Description: The PAGI-SYM Severity index: Heartburn when lying down severity is the participant's assessment of heartburn (burning pain rising in your chest or throat) when lying down over the past 24 hours, where 0=none, 1=very mild, 2=mild, 3=moderate, 4=severe, and 5=very severe. The range of scores is 0 to 5, where higher scores are considered a worse outcome. The outcome measure, change from baseline in Heartburn When Lying Down severity, has a possible range from -5 to +5, with negative values indicating a better outcome (improvement) and positive values indicating a worse outcome.
Time Frame: 4 weeks
Population: The smaller number of participants analyzed is due to missing data at the 4-week follow-up visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aprepitant | Aprepitant-placebo
Number analyzed (Participants) | 56 | 61
units on a scale | -1.2 (1.5) | -0.7 (1.4)
Statistical Analysis 1: Comparison: Aprepitant vs Aprepitant-placebo; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.06, ANCOVA; Mean Difference (Net) = -0.4, 95% CI 2-sided [-0.9 to 0.0]

54. Secondary Outcome: PAGI-SYM Severity Index: Chest Discomfort During the Day Severity
Description: The PAGI-SYM Severity index: Chest discomfort during the day severity is the participant's assessment of feeling of discomfort inside the chest during the day over the past 24 hours, where 0=none, 1=very mild, 2=mild, 3=moderate, 4=severe, and 5=very severe. The range of scores is 0 to 5, where higher scores are considered a worse outcome. The outcome measure, change from baseline in Chest Discomfort During the Day severity, has a possible range from -5 to +5, with negative values indicating a better outcome (improvement) and positive values indicating a worse outcome.
Time Frame: 4 weeks
Population: The smaller number of participants analyzed is due to missing data at the 4-week follow-up visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aprepitant | Aprepitant-placebo
Number analyzed (Participants) | 56 | 61
units on a scale | -1.1 (1.5) | -0.7 (1.4)
Statistical Analysis 1: Comparison: Aprepitant vs Aprepitant-placebo; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.09, ANCOVA; Mean Difference (Net) = -0.4, 95% CI 2-sided [-0.8 to 0.1]

55. Secondary Outcome: PAGI-SYM Severity Index: Chest Discomfort During Sleep Time Severity
Description: The PAGI-SYM Severity index: Chest discomfort during sleep severity is the participant's assessment of feeling of discomfort inside the chest at night (during sleep time) over the past 24 hours, where 0=none, 1=very mild, 2=mild, 3=moderate, 4=severe, and 5=very severe. The range of scores is 0 to 5, where higher scores are considered a worse outcome. The outcome measure, change from baseline in Chest Discomfort During Sleep Time severity, has a possible range from -5 to +5, with negative values indicating a better outcome (improvement) and positive values indicating a worse outcome.
Time Frame: 4 weeks
Population: The smaller number of participants analyzed is due to missing data at the 4-week follow-up visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aprepitant | Aprepitant-placebo
Number analyzed (Participants) | 56 | 61
units on a scale | -0.9 (1.5) | -0.6 (1.4)
Statistical Analysis 1: Comparison: Aprepitant vs Aprepitant-placebo; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.17, ANCOVA; Mean Difference (Net) = -0.3, 95% CI 2-sided [-7 to 0.1]

56. Secondary Outcome: PAGI-SYM Severity Index: Regurgitation During the Day Severity
Description: The PAGI-SYM Severity index: Regurgitation during the day severity is the participant's assessment of regurgitation or reflux (fluid or liquid from your stomach coming up into throat) during the day over the past 24 hours, where 0=none, 1=very mild, 2=mild, 3=moderate, 4=severe, and 5=very severe. The range of scores is 0 to 5, where higher scores are considered a worse outcome. The outcome measure, change from baseline in Regurgitation During the Day severity, has a possible range from -5 to +5, with negative values indicating a better outcome (improvement) and positive values indicating a worse outcome.
Time Frame: 4 weeks
Population: The smaller number of participants analyzed is due to missing data at the 4-week follow-up visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aprepitant | Aprepitant-placebo
Number analyzed (Participants) | 56 | 61
units on a scale | -1.2 (1.7) | -0.5 (1.5)
Statistical Analysis 1: Comparison: Aprepitant vs Aprepitant-placebo; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.009, ANCOVA; Mean Difference (Net) = -0.6, 95% CI 2-sided [-1.1 to -0.2]

57. Secondary Outcome: PAGI-SYM Severity Index: Regurgitation When Lying Down Severity
Description: The PAGI-SYM Severity index: Regurgitation when lying down severity is the participant's assessment of regurgitation or reflux (fluid or liquid from your stomach coming up into throat) when lying down over the past 24 hours, where 0=none, 1=very mild, 2=mild, 3=moderate, 4=severe, and 5=very severe. The range of scores is 0 to 5, where higher scores are considered a worse outcome. The outcome measure, change from baseline in Regurgitation When Lying Down severity, has a possible range from -5 to +5, with negative values indicating a better outcome (improvement) and positive values indicating a worse outcome.
Time Frame: 4 weeks
Population: The smaller number of participants analyzed is due to missing data at the 4-week follow-up visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aprepitant | Aprepitant-placebo
Number analyzed (Participants) | 56 | 61
units on a scale | -1.3 (1.7) | -0.5 (1.3)
Statistical Analysis 1: Comparison: Aprepitant vs Aprepitant-placebo; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.004, ANCOVA; Mean Difference (Net) = -0.7, 95% CI 2-sided [-1.2 to -0.2]

58. Secondary Outcome: PAGI-SYM Severity: Bitter Taste Severity
Description: The PAGI-SYM Severity index: Bitter Taste severity is the participant's assessment of bitter, acid, or sour taste in mouth during the past 24 hours, where 0=none, 1=very mild, 2=mild, 3=moderate, 4=severe, and 5=very severe. The range of scores is 0 to 5, where higher scores are considered a worse outcome. The outcome measure, change from baseline in Bitter Taste Severity score, has a possible range from -5 to +5, with negative values indicating a better outcome (improvement) and positive values indicating a worse outcome.
Time Frame: 4 weeks
Population: The smaller number of participants analyzed is due to missing data at the 4-week follow-up visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aprepitant | Aprepitant-placebo
Number analyzed (Participants) | 56 | 61
units on a scale | -0.8 (1.6) | -0.5 (1.3)
Statistical Analysis 1: Comparison: Aprepitant vs Aprepitant-placebo; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.10, ANCOVA; Mean Difference (Net) = -0.4, 95% CI 2-sided [-0.8 to 0.1]

59. Secondary Outcome: PAGI-SYM Severity Index: Constipation Severity
Description: The PAGI-SYM Severity index: Constipation severity is the participant's assessment of constipation during the past 24 hours, where 0=none, 1=very mild, 2=mild, 3=moderate, 4=severe, and 5=very severe. The range of scores is 0 to 5, where higher scores are considered a worse outcome. The outcome measure, change from baseline in Constipation Severity score, has a possible range from -5 to +5, with negative values indicating a better outcome (improvement) and positive values indicating a worse outcome.
Time Frame: 4 weeks
Population: The smaller number of participants analyzed is due to missing data at the 4-week follow-up visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aprepitant | Aprepitant-placebo
Number analyzed (Participants) | 56 | 61
units on a scale | -0.8 (1.6) | -0.3 (1.5)
Statistical Analysis 1: Comparison: Aprepitant vs Aprepitant-placebo; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.13, ANCOVA; Mean Difference (Net) = -0.4, 95% CI 2-sided [-0.9 to 0.1]

60. Secondary Outcome: PAGI-SYM Severity Index: Diarrhea Severity
Description: The PAGI-SYM Severity index: Diarrhea severity is the participant's assessment of constipation during the past 24 hours, where 0=none, 1=very mild, 2=mild, 3=moderate, 4=severe, and 5=very severe. The range of scores is 0 to 5, where higher scores are considered a worse outcome. The outcome measure, change from baseline in Diarrhea Severity score, has a possible range from -5 to +5, with negative values indicating a better outcome (improvement) and positive values indicating a worse outcome.
Time Frame: 4 weeks
Population: The smaller number of participants analyzed is due to missing data at the 4-week follow-up visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aprepitant | Aprepitant-placebo
Number analyzed (Participants) | 56 | 61
units on a scale | -0.1 (1.4) | -0.2 (1.3)
Statistical Analysis 1: Comparison: Aprepitant vs Aprepitant-placebo; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.98, ANCOVA; Mean Difference (Net) = -0.01, 95% CI 2-sided [-0.5 to 0.4]

61. Secondary Outcome: Gastrointestinal Symptom Rating Scale (GSRS): Total Score
Description: The Gastrointestinal Symptom Rating Scale (GSRS) is a 15-item questionnaire for participants with gastrointestinal discomfort. The GSRS Total Score is the average of the 15 items. Each item is rated on a 0 to 7 scale, where 0 indicates no discomfort and 7 indicates very severe discomfort. The range of scores is 0 to 7, where higher scores are considered a worse outcome.The outcome measure, change from baseline in GSRS Total Score, has a possible range from -7 to +7, with negative values indicating a better outcome (improvement) and positive values indicating a worse outcome.
Time Frame: 4 weeks
Population: The smaller number of participants analyzed is due to missing data at the 4-week follow-up visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aprepitant | Aprepitant-placebo
Number analyzed (Participants) | 56 | 61
units on a scale | -0.8 (0.9) | -0.5 (0.9)
Statistical Analysis 1: Comparison: Aprepitant vs Aprepitant-placebo; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.007, ANCOVA; Mean Difference (Net) = -0.4, 95% CI 2-sided [-0.7 to 0.1]

62. Secondary Outcome: Gastrointestinal Symptom Rating Scale (GSRS): Reflux Score
Description: The Gastrointestinal Symptom Rating Scale (GSRS) is a 15-item questionnaire for participants with gastrointestinal discomfort. The GSRS Reflux Score is a measure of how bothered the participant has been by acid reflux during the past week. The range of scores is 0 to 7, where 0 indicates no discomfort and 7 indicates very severe discomfort. Higher scores are considered a worse outcome.The outcome measure, change from baseline in GSRS Reflux Score, has a possible range from -7 to +7, with negative values indicating a better outcome (improvement) and positive values indicating a worse outcome.
Time Frame: 4 weeks
Population: The smaller number of participants analyzed is due to missing data at the 4-week follow-up visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aprepitant | Aprepitant-placebo
Number analyzed (Participants) | 56 | 61
units on a scale | -1.1 (1.5) | -0.7 (1.6)
Statistical Analysis 1: Comparison: Aprepitant vs Aprepitant-placebo; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.06, ANCOVA; Mean Difference (Net) = -0.5, 95% CI 2-sided [-0.9 to 0.0]

63. Secondary Outcome: Gastrointestinal Symptom Rating Scale (GSRS): Abdominal Pain Score
Description: The Gastrointestinal Symptom Rating Scale (GSRS) is a 15-item questionnaire for participants with gastrointestinal discomfort. The GSRS Abdominal Pain Score is a measure of how bothered the participant has been by pain or discomfort in the upper abdomen or pit of the stomach during the past week. The range of scores is 0 to 7, where 0 indicates no discomfort and 7 indicates very severe discomfort. Higher scores are considered a worse outcome.The outcome measure, change from baseline in GSRS Abdominal Pain Score, has a possible range from -7 to +7, with negative values indicating a better outcome (improvement) and positive values indicating a worse outcome.
Time Frame: 4 week
Population: The smaller number of participants analyzed is due to missing data at the 4-week follow-up visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aprepitant | Aprepitant-placebo
Number analyzed (Participants) | 56 | 61
units on a scale | -1.3 (1.1) | -0.7 (1.0)
Statistical Analysis 1: Comparison: Aprepitant vs Aprepitant-placebo; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.001, ANCOVA; Mean Difference (Net) = -0.6, 95% CI 2-sided [-1.0 to -0.2]

64. Secondary Outcome: Gastrointestinal Symptom Rating Scale (GSRS): Indigestion Score
Description: The Gastrointestinal Symptom Rating Scale (GSRS) is a 15-item questionnaire for participants with gastrointestinal discomfort. The GSRS Indigestion Score is a measure of how bothered the participant has been by indigestion during the past week. The range of scores is 0 to 7, where 0 indicates no discomfort and 7 indicates very severe discomfort. Higher scores are considered a worse outcome.The outcome measure, change from baseline in GSRS Indigestion Score, has a possible range from -7 to +7, with negative values indicating a better outcome (improvement) and positive values indicating a worse outcome.
Time Frame: 4 weeks
Population: The small number of participants analyzed is due to missing data at the 4-week follow-up visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aprepitant | Aprepitant-placebo
Number analyzed (Participants) | 56 | 61
units on a scale | -0.7 (1.3) | -0.7 (1.1)
Statistical Analysis 1: Comparison: Aprepitant vs Aprepitant-placebo; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.28, ANCOVA; Mean Difference (Net) = -0.2, 95% CI 2-sided [-0.6 to 0.2]

65. Secondary Outcome: Gastrointestinal Symptom Rating Scale (GSRS): Diarrhea Score
Description: The Gastrointestinal Symptom Rating Scale (GSRS) is a 15-item questionnaire for participants with gastrointestinal discomfort. The GSRS Diarrhea Score is a measure of how bothered the participant has been by diarrhea during the past week. The range of scores is 0 to 7, where 0 indicates no discomfort and 7 indicates very severe discomfort. Higher scores are considered a worse outcome.The outcome measure, change from baseline in GSRS Diarrhea Score, has a possible range from -7 to +7, with negative values indicating a better outcome (improvement) and positive values indicating a worse outcome.
Time Frame: 4 weeks
Population: The smaller number of participants analyzed is due to missing data at the 4-week follow-up visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aprepitant | Aprepitant-placebo
Number analyzed (Participants) | 56 | 61
units on a scale | -0.5 (1.6) | 0.1 (1.3)
Statistical Analysis 1: Comparison: Aprepitant vs Aprepitant-placebo; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.05, ANCOVA; Mean Difference (Net) = -0.5, 95% CI 2-sided [-1.0 to 0.0]

66. Secondary Outcome: Gastrointestinal Symptom Rating Scale (GSRS): Constipation Score
Description: The Gastrointestinal Symptom Rating Scale (GSRS) is a 15-item questionnaire for participants with gastrointestinal discomfort. The GSRS Constipation Score is a measure of how bothered the participant has been by constipation during the past week. The range of scores is 0 to 7, where 0 indicates no discomfort and 7 indicates very severe discomfort. Higher scores are considered a worse outcome.The outcome measure, change from baseline in GSRS Constipation Score, has a possible range from -7 to +7, with negative values indicating a better outcome (improvement) and positive values indicating a worse outcome.
Time Frame: 4 weeks
Population: The smaller number of participants analyzed is due to missing data at the 4-week follow-up visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aprepitant | Aprepitant-placebo
Number analyzed (Participants) | 56 | 61
units on a scale | -0.8 (1.3) | -0.4 (1.5)
Statistical Analysis 1: Comparison: Aprepitant vs Aprepitant-placebo; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.08, ANCOVA; Mean Difference (Net) = -0.4, 95% CI 2-sided [-0.9 to 0.1]

67. Secondary Outcome: Brief Pain Inventory: Severity Score
Description: The Brief Pain Inventory: Severity Score is the average of four questions in which the participant rates his or her pain: the worse pain in the past 24 hours, the least pain in the past 24 hours, average pain, and pain right now. The range of possible scores is 0 to 10, with higher scores indicating more severe pain. The outcome measure, change from baseline in Brief Pain Inventory Severity Score, has a possible range from -10 to +10, with negative values indicating a better outcome (improvement) and positive values indicating a worse outcome.
Time Frame: 4 weeks
Population: The smaller number of participants analyzed is due to missing data at the 4-week follow-up visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aprepitant | Aprepitant-placebo
Number analyzed (Participants) | 56 | 61
units on a scale | -1.0 (2.6) | -0.7 (2.3)
Statistical Analysis 1: Comparison: Aprepitant vs Aprepitant-placebo; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.53, ANCOVA; Mean Difference (Net) = -0.3, 95% CI 2-sided [-1.1 to 0.6]

68. Secondary Outcome: Brief Pain Inventory: Interference Score
Description: The Brief Pain Inventory: Interference Score is the average of seven questions in which the participant rates the degree to which his or her pain interferes with daily functions and mood: general activity, mood, walking ability, normal work, relationships, sleep, enjoyment of life. The range of possible scores is 0 to 10, with higher scores indicating more interference caused by pain. The outcome measure, change from baseline in Brief Pain Inventory Interference Score, has a possible range from -10 to +10, with negative values indicating a better outcome (improvement) and positive values indicating a worse outcome.
Time Frame: 4 weeks
Population: The smaller number of participants analyzed is due to missing data at the 4-week follow-up visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aprepitant | Aprepitant-placebo
Number analyzed (Participants) | 56 | 61
units on a scale | -1.1 (2.6) | -1.0 (2.6)
Statistical Analysis 1: Comparison: Aprepitant vs Aprepitant-placebo; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.38, ANCOVA; Mean Difference (Net) = -0.4, 95% CI 2-sided [-1.3 to 0.5]

69. Secondary Outcome: Beck Depression Inventory (BDI) Score
Description: The Beck Depression Inventory (BDI) survey is comprised of 21 multiple choice questions that relate to depression, cognition, and physical well-being and is used to quantify depression. The BDI total score is the sum of the 21 items, where each item ranges from 0 to 3 (lower scores are less severe, higher scores are more severe). The range for the BDI total score is 0 to 63, where lower scores indicate less depression and higher scores indicate more severe depression. The outcome measure, change from baseline in BDI score, has a possible range from -63 to +63, with negative values indicating a better outcome (improvement) and positive values indicating a worse outcome.
Time Frame: 4 weeks
Population: The smaller number of participants analyzed is due to missing data at the 4-week follow-up visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aprepitant | Aprepitant-placebo
Number analyzed (Participants) | 56 | 61
units on a scale | -4.6 (8.5) | -2.4 (5.9)
Statistical Analysis 1: Comparison: Aprepitant vs Aprepitant-placebo; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.09, ANCOVA; Mean Difference (Net) = -2.2, 95% CI 2-sided [-4.7 to 0.4]

70. Secondary Outcome: State-Trait Anxiety Inventory (STAI): State Anxiety Score
Description: The State-Trait Anxiety Inventory (STAI): State anxiety score is the sum of scores from 20 questions relating to state anxiety, which is a temporary state varying in intensity. The possible range of scores is from 20 to 80, with increasing scores considered a worse outcome. The outcome measure, change from baseline in STAI State Anxiety score, has a possible range from -60 to +60, with negative values indicating a better outcome (improvement) and positive values indicating a worse outcome.
Time Frame: 4 weeks
Population: The smaller number of participants analyzed is due to missing data at the 4-week follow-up visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aprepitant | Aprepitant-placebo
Number analyzed (Participants) | 56 | 61
units on a scale | -3.1 (8.7) | -1.7 (10.6)
Statistical Analysis 1: Comparison: Aprepitant vs Aprepitant-placebo; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.28, ANCOVA; Mean Difference (Net) = -1.8, 95% CI 2-sided [-5.2 to 1.5]

71. Secondary Outcome: State-Trait Anxiety Inventory (STAI): Trait Anxiety Score
Description: The State-Trait Anxiety Inventory (STAI): Trait anxiety score is the sum of scores from 20 questions pertaining to trait anxiety, which is a general propensity to be anxious. The possible range of scores is from 20 to 80, with increasing scores considered a worse outcome. The outcome measure, change from baseline in STAI Trait Anxiety score, has a possible range from -60 to +60, with negative values indicating a better outcome (improvement) and positive values indicating a worse outcome.
Time Frame: 4 weeks
Population: The smaller number of participants analyzed is due to missing data at the 4-week follow-up visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aprepitant | Aprepitant-placebo
Number analyzed (Participants) | 56 | 61
units on a scale | -1.8 (8.8) | -0.7 (8.4)
Statistical Analysis 1: Comparison: Aprepitant vs Aprepitant-placebo; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.30, ANCOVA; Mean Difference (Net) = -1.6, 95% CI 2-sided [-4.6 to 1.4]

72. Secondary Outcome: Satiety Test, Volume Consumed
Description: The Satiety Test measures the total volume of liquid (Ensure) that the participant is able to consume. The participant drinks 150 mL of Ensure every 5 minutes until he/she is completely full. The outcome measure is the change from baseline in volume of liquid (Ensure) consumed (mL), where positive values indicate a positive outcome (improvement).
Time Frame: 4 weeks
Population: The smaller number of participants analyzed is due to missing data at the 4-week follow-up visit.
Measure: Median (Inter-Quartile Range); unit: mL
Arm/Group | Aprepitant | Aprepitant-placebo
Number analyzed (Participants) | 48 | 55
mL | -13.0 [-75.85 to 49.85] | 9.2 [-56.35 to 74.75]
Statistical Analysis 1: Comparison: Aprepitant vs Aprepitant-placebo; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.40, ANCOVA; Mean Difference (Net) = -21.2, 95% CI 2-sided [-70.5 to 28.1]

73. Secondary Outcome: Electrogastrography (EGG): Bradygastria (1-<2.5 Cpm) at 4 Weeks, Baseline Measurement
Description: Electrogastrography (EGG) is a test which records the electrical pacemaking signals that travel through the stomach muscles and control the muscles' contractions. Normal pacing is considered 2.5-3.7 cycles per minute (cpm). Bradygastria is when the rate of electrical activity in the stomach is <2.5 cycles per minute for at least 1 minute (a decrease in electrical activity in the stomach). The average power in frequency region is the percentage of time that the dominant EGG frequencies are in a given frequency: bradygastria, normal, tachygastria, or duodenal. The outcome measure is the change from baseline (here, baseline refers to the test performed during screening, not the baseline value of the EGG test) in percent of time with frequencies in the ranges, where negative values for bradygastria indicate improvement (less time in a dysrhythmic state).
Time Frame: 4 weeks
Population: The smaller number of participants analyzed is due to missing data at the 4-week follow-up visit.
Measure: Mean (Standard Deviation); unit: average power in frequency region, %
Arm/Group | Aprepitant | Aprepitant-placebo
Number analyzed (Participants) | 48 | 55
average power in frequency region, % | -4.6 (24.6) | 2.8 (21.5)
Statistical Analysis 1: Comparison: Aprepitant vs Aprepitant-placebo; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.28, ANCOVA; Mean Difference (Net) = -4.2, 95% CI 2-sided [-12.0 to 3.5]

74. Secondary Outcome: Electrogastrography (EGG): Bradygastria (1-<2.5 Cpm) at 4 Weeks, 0-30 Post-satiety Measurement
Description: Electrogastrography (EGG) is a test which records the electrical pacemaking signals that travel through the stomach muscles and control the muscles' contractions. The 0-30 post-satiety measurement of the test is that taken 30 minutes after the participant consumes Ensure until feeling completely full. Normal pacing is considered 2.5-3.7 cycles per minute (cpm). Bradygastria is when the rate of electrical activity in the stomach is <2.5 cycles per minute for at least 1 minute. Average power in frequency region is the % of time that the dominant EGG frequencies are in a given frequency: bradygastria, normal, tachygastria, or duodenal. The outcome measure is the change from baseline (baseline refers to test performed during screening, not baseline value of the EGG test) in % of time with frequencies in the ranges. Negative values for bradygastria indicate improvement (less time in a dysrhythmic state).
Time Frame: 4 weeks
Population: The smaller number of participants analyzed is due to missing data at the 4-week follow-up visit.
Measure: Mean (Standard Deviation); unit: average power in frequency region, %
Arm/Group | Aprepitant | Aprepitant-placebo
Number analyzed (Participants) | 48 | 55
average power in frequency region, % | 2.1 (17.7) | 0.5 (19.4)
Statistical Analysis 1: Comparison: Aprepitant vs Aprepitant-placebo; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.47, ANCOVA; Mean Difference (Net) = 2.4, 95% CI 2-sided [-4.1 to 8.9]

75. Secondary Outcome: Electrogastrography (EGG): Normogastria (2.5-<3.8 Cpm) at 4 Weeks, Baseline Measurement
Description: Electrogastrography (EGG) is a test which records the electrical pacemaking signals that travel through the stomach muscles and control the muscles' contractions. Normal pacing (normogastria) is considered 2.5-3.7 cycles per minute (cpm). The average power in frequency region is the percentage of time that the dominant EGG frequencies are in a given frequency: bradygastria, normal, tachygastria, or duodenal. The outcome measure is the change from baseline (here, baseline refers to the test performed during screening, not the baseline value of the EGG test) in percent of time with frequencies in the ranges, where positive values for normal rates indicate an increase in the normal pacing (improvement).
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: average power in frequency region, %
Arm/Group | Aprepitant | Aprepitant-placebo
Number analyzed (Participants) | 48 | 55
average power in frequency region, % | 1.0 (19.9) | -1.0 (16.5)
Statistical Analysis 1: Comparison: Aprepitant vs Aprepitant-placebo; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.68, ANCOVA; Mean Difference (Net) = 1.2, 95% CI 2-sided [-4.5 to 6.9]

76. Secondary Outcome: Electrogastrography (EGG): Normogastria (2.5-<3.8 Cpm) at 4 Weeks, 0-30 Post-satiety Measurement
Description: Electrogastrography (EGG) is a test which records the electrical pacemaking signals that travel through the stomach muscles and control the muscles' contractions. The 0-30 post-satiety measurement that taken 30 minutes after the participant consumes Ensure until feeling completely full. Normal pacing (normogastria) is considered 2.5-3.7 cycles per minute (cpm). The average power in frequency region is the percentage of time that the dominant EGG frequencies are in a given frequency: bradygastria, normal, tachygastria, or duodenal. The outcome measure is the change from baseline (baseline refers to the test performed during screening, not the baseline value of the EGG test) in percent of time with frequencies in the ranges, where positive values for normal rates indicate an increase in the normal pacing (improvement).
Time Frame: 4 weeks
Population: The smaller number of participants analyzed is due to missing data at the 4-week follow-up visit.
Measure: Mean (Standard Deviation); unit: average power in frequency region, %
Arm/Group | Aprepitant | Aprepitant-placebo
Number analyzed (Participants) | 48 | 55
average power in frequency region, % | 1.0 (15.8) | 0.8 (15.1)
Statistical Analysis 1: Comparison: Aprepitant vs Aprepitant-placebo; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.48, ANCOVA; Mean Difference (Net) = 2.0, 95% CI 2-sided [-3.6 to 7.6]

77. Secondary Outcome: Electrogastrography (EGG): Tachygastria (3.8-10 Cpm) at 4 Weeks, Baseline Measurement
Description: Electrogastrography (EGG) is a test which records the electrical pacemaking signals that travel through the stomach muscles and control the muscles' contractions. Normal pacing is considered 2.5-3.7 cycles per minute (cpm). Tachygastria is when the rate of electrical activity in the stomach is 3.8-10 cycles per minute for at least 1 minute (an increase in electrical activity in the stomach). The average power in frequency region is the percentage of time that the dominant EGG frequencies are in a given frequency: bradygastria, normal, tachygastria, or duodenal. The outcome measure is the change from baseline (here, baseline refers to the test performed during screening, not the baseline value of the EGG test) in percent of time with frequencies in the ranges, where negative values for tachygastria indicate improvement (less time in a dysrhythmic state).
Time Frame: 4 weeks
Population: The smaller number of participants analyzed is due to missing data at the 4-week follow-up visit.
Measure: Mean (Standard Deviation); unit: average power in frequency region, %
Arm/Group | Aprepitant | Aprepitant-placebo
Number analyzed (Participants) | 48 | 55
average power in frequency region, % | 1.5 (12.3) | -1.6 (12.0)
Statistical Analysis 1: Comparison: Aprepitant vs Aprepitant-placebo; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.43, ANCOVA; Mean Difference (Net) = 1.5, 95% CI 2-sided [-2.2 to 5.1]

78. Secondary Outcome: Electrogastrography (EGG): Tachygastria (3.8-10 Cpm) at 4 Weeks, 0-30 Post-satiety Measurement
Description: Electrogastrography (EGG) is a test which records the electrical pacemaking signals that travel through the stomach muscles and control the muscles' contractions. The 0-30 post-satiety measurement that taken 30 minutes after the participant consumes Ensure until feeling completely full. Normal pacing is considered 2.5-3.7 cycles per minute (cpm). Tachygastria is when the rate of electrical activity in the stomach is 3.8-10 cycles per minute for at least 1 minute (an increase in electrical activity in the stomach). The average power in frequency region is the percentage of time that the dominant EGG frequencies are in a given frequency: bradygastria, normal, tachygastria, or duodenal. The outcome measure is the change from baseline (here, baseline refers to the test performed during screening, not the baseline value of the EGG test) in percent of time with frequencies in the ranges, where negative values for tachygastria indicate improvement (less time in a dysrhythmic state).
Time Frame: 4 weeks
Population: The smaller number of participants analyzed is due to missing data at the 4-week follow-up visit.
Measure: Mean (Standard Deviation); unit: average power in frequency region, %
Arm/Group | Aprepitant | Aprepitant-placebo
Number analyzed (Participants) | 48 | 55
average power in frequency region, % | -2.1 (9.7) | -0.8 (14.1)
Statistical Analysis 1: Comparison: Aprepitant vs Aprepitant-placebo; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.01, ANCOVA; Mean Difference (Net) = -4.8, 95% CI 2-sided [-8.5 to -1.2]

79. Secondary Outcome: Electrogastrography (EGG): Duodenal (>10-15 Cpm) at 4 Weeks, Baseline Measurement
Description: Electrogastrography (EGG) is a test which records the electrical pacemaking signals that travel through the stomach muscles and control the muscles' contractions. Normal pacing is considered 2.5-3.7 cycles per minute (cpm). Duodenal is when the rate of electrical activity in the stomach is >10-15 cycles per minute for at least 1 minute. The average power in frequency region is the percentage of time that the dominant EGG frequencies are in a given frequency: bradygastria, normal, tachygastria, or duodenal. The outcome measure is the change from baseline (here, baseline refers to the test performed during screening, not the baseline value of the EGG test) in percent of time with frequencies in the ranges, where negative values for duodenal indicate improvement (less time in a dysrhythmic state).
Time Frame: 4 weeks
Population: The smaller number of participants analyzed is due to missing data at the 4-week followup visit.
Measure: Mean (Standard Deviation); unit: average power in frequency region, %
Arm/Group | Aprepitant | Aprepitant-placebo
Number analyzed (Participants) | 48 | 55
average power in frequency region, % | 2.1 (13.5) | -0.2 (13.4)
Statistical Analysis 1: Comparison: Aprepitant vs Aprepitant-placebo; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.57, ANCOVA; Mean Difference (Net) = 1.4, 95% CI 2-sided [-3.4 to 6.1]

80. Secondary Outcome: Electrogastrography (EGG): Duodenal (>10-15 Cpm) at 4 Weeks, 0-30 Post-satiety Measurement
Description: Electrogastrography (EGG) is a test which records the electrical pacemaking signals that travel through the stomach muscles and control the muscles' contractions. The 0-30 post-satiety measurement that taken 30 minutes after the participant consumes Ensure until feeling completely full. Normal pacing is considered 2.5-3.7 cycles per minute (cpm). Duodenal is when the rate of electrical activity in the stomach is >10-15 cycles per minute for at least 1 minute. The average power in frequency region is the percentage of time that the dominant EGG frequencies are in a given frequency: bradygastria, normal, tachygastria, or duodenal. The outcome measure is the change from baseline (here, baseline refers to the test performed during screening, not the baseline value of the EGG test) in percent of time with frequencies in the ranges, where negative values for duodenal indicate improvement (less time in a dysrhythmic state).
Time Frame: 4 weeks
Population: The smaller number of participants analyzed is due to missing data at the 4-week follow-up visit.
Measure: Mean (Standard Deviation); unit: average power in frequency region, %
Arm/Group | Aprepitant | Aprepitant-placebo
Number analyzed (Participants) | 48 | 55
average power in frequency region, % | -0.8 (7.3) | -0.5 (5.5)
Statistical Analysis 1: Comparison: Aprepitant vs Aprepitant-placebo; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.34, ANCOVA; Mean Difference (Net) = -0.84, 95% CI 2-sided [-2.6 to 1.0]

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Aprepitant | Aprepitant-placebo
All-Cause Mortality (participants affected / at risk) | 0/63 | 0/63
Serious Adverse Events (participants affected / at risk) | 1/63 | 0/63
Other Adverse Events (participants affected / at risk) | 21/63 | 11/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aprepitant (N=63) | Aprepitant-placebo (N=63)
Hypoglycemia (Endocrine disorders) | 1 (1) | 0 (0) — The patient was determined to be diabetic and had delayed retention. Hospitalization due to nausea and vomiting.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aprepitant (N=63) | Aprepitant-placebo (N=63)
Nausea, vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flashing lights/floaters (Eye disorders) | 0 (0) | 1 (1)
Bruising (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 2 (2)
Gastrointestinal - Other (abdominal pain) (Gastrointestinal disorders) | 3 (3) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea, abdominal pain, diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diarrhea, syncope (General disorders) | 1 (1) | 0 (0) — Reaction to different medication; not study-related
Musculoskeletal - Other (neck and right hand pain) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Diarrhea, loss of appetite (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal - Other (fainting sensation) (Gastrointestinal disorders) | 1 (1) | 0 (0)
Renal/Genitourinary - Other (Bleeding) (Renal and urinary disorders) | 1 (1) | 0 (0)
Fibromyalgia cystitis (Renal and urinary disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rhinitis (Immune system disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Gastrointestinal - Other (Nausea, malaise) (Gastrointestinal disorders) | 1 (1) | 0 (0)
Musculoskeletal - Other (Limb pain) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nosebleed (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Bruising (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — High blood pressure, shortness of breath, dizziness, palpitations
Depression (Psychiatric disorders) | 0 (0) | 1 (1) — Withdrawal from depression medication caused dizziness, vertigo, and light sensitivity
Neurology - other (Nervous system disorders) | 0 (0) | 1 (1) — Migraines, pain, stiffness, chest pain, heart palpitations, lower left quad pain, chills, fever, burping

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No